

## STATISTICAL ANALYSIS PLAN

**Study Title:** A Phase 3 Randomized, Double-Blind, Placebo-Controlled,

Parallel Group, Multicenter Study Evaluating the Efficacy and Safety of Remdesivir in Participants with Severely Reduced Kidney Function who are Hospitalized for

COVID-19

Name of Test Drug: Remdesivir

Study Number: GS-US-540-5912

**Protocol Version (Date):** Original: 07 December 2020

Amendment 1: 28 January 2021 Amendment 2: 02 August 2021 Amendment 3: 27 August 2021

**Analysis Type:** Final Analysis

**Analysis Plan Version:** SAP v1.0

**Analysis Plan Date:** 22 July 2022

Analysis Plan Author(s): PPD & PPD

CONFIDENTIAL AND PROPRIETARY INFORMATION

# TABLE OF CONTENTS

| ST | ATISTI | CAL ANA | LYSIS PLAN | 1 |
|---|---|---|---|---|
| TA | BLE OI | CONTEN | NTS | 2 |
| LIS | ST OF I | N-TEXT T | ABLES | 4 |
| LIS | ST OF I | N-TEXT F | IGURES | 4 |
| LIS | T OF A | BBREVIA | ATIONS | 5 |
| 1. | INTRODUCTION | | | 7 |
| | 1.1. | Study Objectives | | |
| | 1.2. | The second secon | esign | |
| | 1.3. | | Size and Power | |
| 2. | | | | |
| | 2.1. | 2.1. Interim Analyses | | |
| | 2.2. | | | |
| | 2.3. | | nalysis | |
| | 2.4. | | from Protocol-Specified Analyses | |
| 3. | GENI | | NSIDERATIONS FOR DATA ANALYSES | |
| | 3.1. | | s Sets | |
| | 3.1. | 3.1.1. | All Randomized Analysis Set. | |
| | | 3.1.2. | Full Analysis Set | |
| | | 3.1.3. | Safety Analysis Set | |
| | | CCI | Salety Filmly do See | |
| | 3.2. | Participa | ant Grouping | 12 |
| | 3.3. | | | |
| | 3.4. | | | 13 |
| | 3.5. | Multiple | e Comparisons | 13 |
| | 3.6. | | | 14 |
| | | 3.6.1. | Missing Data | 14 |
| | | 3.6.2. | Outliers | |
| | 3.7. | Data Ha | ndling Conventions and Transformations | 14 |
| | 3.8. | Analysis | s Visit Windows | 16 |
| | | 3.8.1. | Definition of Study Day | |
| | | 3.8.2. | Analysis Visit Windows | 16 |
| | | 3.8.3. | Selection of Data in the Event of Multiple Records in an Analysis Visit | |
| | | | Window | |
| | 3.9. | Change | from Protocol-Specified General Considerations | 19 |
| 4. | PARTICIPANT DISPOSITION | | | |
| | 4.1. | Participant Enrollment and Disposition. | | |
| | 4.2. | | | 21 |
| | 4.3. | 4.3. Protocol Deviations | | 21 |
| 5. | BASE | BASELINE CHARACTERISTICS | | |
| | 5.1. | 5.1. Demographics and Baseline Characteristics | | |
| | 5.2. | | | |
| | 5.3. | | History | |

| 6. | EFFI | CACY AN | ALYSES | | 24 |
|---|---|---|---|---|---|
| | 6.1. | Primary Efficacy Endpoint | | | 24 |
| | | 6.1.1. | | ficacy Endpoint | |
| | | 6.1.2. | | Primary Efficacy Endpoint | |
| | | 6.1.3. | | nary Efficacy Endpoint | |
| | | 6.1.4. | | rimary Efficacy Endpoint | |
| | 6.2. | | | | |
| | CCI | 6.2.1. | Analysis of Secondary Effica | ncy Endpoints | 25 |
| | CCI | ÷ ā | | | |
| | 6.4. | Changes | from Protocol-Specified Effica | cy Analyses | 29 |
| 7. | SAFETY ANALYSES | | | | 30 |
| | 7.1. | Adverse | Events and Deaths | | 30 |
| | | 7.1.1. | Adverse Event Dictionary | | 30 |
| | | 7.1.2. | Adverse Event Severity | | 30 |
| | | 7.1.3. | Relationship of Adverse Eve | nts to Study Drug | 30 |
| | | 7.1.4. | Serious Adverse Events | | 30 |
| | | 7.1.5. | Treatment-Emergent Advers | e Events | 30 |
| | | | 7.1.5.1. Definition of T | reatment-Emergent Adverse Events | 30 |
| | | | 7.1.5.2. Incomplete Date | es | 31 |
| | | 7.1.6. | Summaries of Adverse Even | ts and Deaths | 31 |
| | 7.2. | | | 32 | |
| | | 7.2.1. | Summaries of Numeric Labo | ratory Results | 33 |
| | | 7.2.2. | Graded Laboratory Values | | 34 |
| | | | 7.2.2.1. Treatment-Eme | ergent Laboratory Abnormalities | 34 |
| | | | 7.2.2.2. Summaries of l | Laboratory Abnormalities | 34 |
| | | 7.2.3. | Liver-Related Laboratory Ev | aluations | 35 |
| | 7.3. Vital Signs and Respiratory Status | | | 35 | |
| | 7.4. | 4. Concomitant Medications | | | 36 |
| | 7.5. | Other Safety Measures | | | 36 |
| | 7.6. Changes from Protocol-Specified Safety Analyses | | | 36 | |
| CCI | | | | | |
| | | 0 | | | |
| 9. | REFE | ERENCES | | | 39 |
| 10. | | | | | |
| | | NDICES | | | 41 |
| | APPE | THE PARTY | | | 4/ |

# LIST OF IN-TEXT TABLES

| Table 3-1. | Analysis Visit Windows for Chemistry (Except for SCr), Hematology, and Coagulation Laboratory Tests | 17 |
|---|---|---|
| CCI<br>Table 3-3. | Analysis Visit Window for 8-Point Ordinal Scale Collected after Day 44 | |
| | LIST OF IN-TEXT FIGURES | |
| Figure 1-1. | Study Schema | 8 |

#### LIST OF ABBREVIATIONS

AE adverse event

AKI acute kidney injury

ALT alanine aminotransferase

AST aspartate aminotransferase

BLQ below the limit of quantitation

BMI body mass index
BUN blood urea nitrogen
CI confidence interval
CKD chronic kidney disease
CMH Cochran-Mantel-Haenszel

CoV coronavirus

COVID-19 coronavirus disease 2019

CRF case report form
CSR clinical study report
DAIDS Division of AIDS

DAVG Time-weighted average change from baseline

DMC data monitoring committee
ED Emergency department
ESKD end-stage kidney disease

ET early termination
FAS Full Analysis Set
Hb Hemoglobin
HLT high-level term

HLGT high-level group term

International Conference on Harmonization (of Technical Requirements for Registration of

Pharmaceuticals for Human Use)

IMV Invasive mechanical ventilation

IV Intravenous

IXRS interactive voice or web response system

LLT lower-level term LOQ limit of quantitation

MedDRA Medical Dictionary for Regulatory Activities

PCR polymerase chain reaction

PK pharmacokinetics
PT preferred term
PTM Placebo to match

Q1, Q3 first quartile, third quartile

RDV remdesivir

RRT renal replacement therapy

SAE serious adverse event SAP statistical analysis plan

SARS severe acute respiratory syndrome SBECD sulfobutylether-beta-cyclodextrin

SCr serum creatinine
SD standard deviation

SI (units) international system of units

SOC system organ class SpO<sub>2</sub> oxygen saturation

TEAE treatment-emergent adverse event

TFLs tables, figures, and listings ULN upper limit of normal

US United States

WHO World Health Organization

## 1. INTRODUCTION

This statistical analysis plan (SAP) describes the statistical analysis methods and data presentations to be used in tables, figures, and listings (TFLs) in the clinical study report (CSR) for Study GS-US-540-5912. This SAP is based on the study protocol Amendment 3 dated 27 August 2021 and the electronic case report form (eCRF). This SAP will be finalized before data finalization and unblinding. Any changes made after the finalization of the SAP will be documented in the CSR.

# 1.1. Study Objectives

The primary objective of this study is as follows:

• To evaluate whether remdesivir (RDV) reduces the composite risk of death or invasive mechanical ventilation (IMV) through Day 29 in participants with severely reduced kidney function who are hospitalized for coronavirus disease 2019 (COVID-19)

The secondary objectives of this study are as follows:

- To evaluate whether RDV reduces the risk of death through Day 29
- To evaluate whether RDV reduces the risk of IMV through Day 29
- To evaluate the time to recovery (defined as satisfying category 1, 2, or 3 by an 8-point ordinal scale)
- To evaluate the effect of RDV on clinical status assessed by an 8-point ordinal scale at Day 15 and Day 29
- To evaluate the effect of RDV on renal replacement therapy (RRT)-free days (among those without end-stage kidney disease [ESKD]) through Day 29
- To evaluate the effect of RDV on recovery through Day 29
- To evaluate the safety and tolerability of RDV in participants with severely reduced kidney function who are hospitalized for COVID-19





# 1.2. Study Design

This is a Phase 3 randomized, double-blind, placebo-controlled, parallel-group, multicenter study evaluating the efficacy and safety of RDV therapy in participants with severely reduced kidney function who are hospitalized for COVID-19.

Figure 1-1. Study Schema



\*Day 60 follow-up phone call

Approximately 1,116 eligible participants are planned to be randomized in a 2:1 ratio to receive RDV or saline as placebo, according to the following treatment regimen, in addition to standard of care therapy:

**Treatment Group A (N = 744)**: IV RDV 200 mg on Day 1 followed by IV RDV 100 mg once daily from Day 2 up to Day 5

**Treatment Group B (N = 372)**: IV saline as placebo on Day 1 followed by IV saline as placebo once daily from Day 2 up to Day 5

Randomization will be stratified by:

- ESKD requiring chronic dialysis
- High-flow oxygen requirement
- Region (United States [US] vs. ex-US)

All participants will be requested to continue assessments during study hospitalization and any subsequent re-hospitalization to the same institution during Days 1 through 29 and attend the Day 60 phone follow-up (whether hospitalized or as an outpatient).

The schedule of assessments is provided as an appendix (Appendix 1).

## 1.3. Sample Size and Power

A total of approximately 1116 participants are planned to be randomized in a 2:1 ratio to 2 groups (744 in the RDV group and 372 in the saline as placebo group).

This sample size achieves approximately 85% power to detect a hazard ratio of 0.70 at a two-sided alpha level of 0.05. In the sample size calculation, it is assumed that the event rate in the saline as placebo group is 35%. The hazard ratio and event rate in the saline as placebo group are based on the most conservative estimates of the primary endpoint (composite of all-cause mortality or IMV) and the key  $\alpha$ -controlled secondary endpoint (all-cause mortality) through Day 29 among a subset of participants with eGFR < 60 mL/min in the Division of Microbiology and Infectious Diseases Protocol 20-0006 Adaptive COVID-19 Treatment Trial (ACTT)-1 (hazard ratio of 0.67 and placebo rate of 33%).

The sample size calculation was done using software EAST (Version 6.5, module for log-rank test given accrual duration [120 days] and study duration [149 days] and 1 interim analysis at 50% information fraction using the Lan-Demets approach with O'Brien-Fleming type spending function).

#### 2. TYPE OF PLANNED ANALYSIS

# 2.1. Interim Analyses

Prior to the final analysis, interim analyses may be conducted, and the analyses may be submitted to regulatory agencies to seek guidance for the overall clinical development program.

## 2.2. DMC Analyses

Two formal DMC meetings were planned for this study and were specified in protocol Sections 8.2 and 8.10. The first meeting has occurred and was conducted after the first 100 participants completed the Day 29 assessment. The purpose of this meeting was to review safety data, including renal and hepatic toxicity. The second meeting was planned after 50% of participants completed the Day 29 assessment. The purpose of this meeting was to review safety and provide a formal evaluation of futility and efficacy. However, this analysis was not performed due to the stop of study enrollment prior to reaching 50% of planned enrollment.

In addition to the above mentioned 2 formal DMC analyses, the DMC was provided with blinded safety listings including Grade 3 or higher AEs and SAEs every week for the first 2 weeks after the first participant was enrolled followed by every 2 weeks thereafter.

All details on DMC analyses are documented in the approved DMC charter.

## 2.3. Final Analysis

The final analysis will be performed after all participants have completed or discontinued from the study, outstanding data queries have been resolved or adjudicated as unresolvable, and the data have been cleaned and finalized.

The analysis of the primary endpoint of all-cause mortality or IMV through Day 29 and the key  $\alpha$ -controlled secondary endpoint of all-cause mortality through Day 29 will be conducted at the final analysis (see Section 3.5 for prespecified testing strategy). The overall Type I error rate will be controlled at the two-sided 0.05 significance level.

## 2.4. Change from Protocol-Specified Analyses

The second formal DMC analysis was not performed due to the stop of study enrollment prior to reaching 50% of planned enrollment. The reason for stopping enrollment was that it became clear the study would not fully enroll in a reasonable timeframe even after implementing enrollment mitigation strategies. The decision to stop study enrollment was documented in the 16 December 2021 Study Management Team meeting minutes.

## 3. GENERAL CONSIDERATIONS FOR DATA ANALYSES

Analysis results will be presented using descriptive statistics. For categorical variables, the number and percentage of participants in each category will be presented; for continuous variables, the number of participants (n), mean, standard deviation (SD) or standard error (SE), median, first quartile (Q1), third quartile (Q3), minimum, and maximum will be presented.

By-participant listings will be presented for all participants in the All Randomized Analysis Set and sorted by participant identification (ID) number, visit date, and time (if applicable). Data collected on log forms, such as adverse events (AEs), will be presented in chronological order for each participant. The treatment group to which participants were randomized will be used in the listings. Age, sex at birth, race, and ethnicity will be included in the listings, as space permits.

# 3.1. Analysis Sets

Analysis sets define the participants to be included in an analysis. Analysis sets and their definitions are provided in this section. Participants included in each analysis set will be determined before the study blind is broken for analysis. The analysis set will be identified and included as a subtitle of each table, figure, and listing.

For each analysis set, the number and percentage of participants eligible for inclusion will be summarized by treatment group.

A listing of reasons for exclusion from analysis sets will be provided by participant.

#### CCI

#### 3.1.1. All Randomized Analysis Set

All Randomized Analysis Set includes all participants who were randomized in the study.

## 3.1.2. Full Analysis Set

The primary analysis set for efficacy analysis is defined as the Full Analysis Set (FAS), which will include all participants who (1) are randomized into the study, and (2) have received at least 1 dose of study drug.

#### 3.1.3. Safety Analysis Set

The primary analysis set for safety analyses is defined as the Safety Analysis Set, which will include all participants who (1) are randomized into the study and (2) have received at least 1 dose of study drug.



#### 3.1.7. Virology Analysis Set

The Virology Analysis Set will include all participants who (1) are randomized into the study, (2) have received at least 1 dose of RDV, and (3) have positive SARS-CoV-2 viral load at baseline (a result of "No SARS-CoV-2 detected" is considered as negative, results of Inconclusive, < limit of quantitation (LOQ) SARSCoV2 detected, and numerical results are considered as positive).

# 3.2. Participant Grouping

For analyses based on the All Randomized Analysis Set and FAS, participants will be grouped according to the treatment to which they were randomized. For analyses based on Safety Analysis Set. CCI Virology Analysis Set and CCI participants will be grouped according to the actual treatment they received.

The actual treatment received will differ from the randomized treatment only when their actual treatment differs from randomized treatment for the entire treatment duration.

#### 3.3. Strata and Covariates

Participants will be randomly assigned to treatment groups via the interactive voice or web response system (IXRS) in a 2:1 ratio using a stratified randomization schedule. Randomization will be stratified by:

- ESKD requiring chronic dialysis (Yes, No)
- High-flow oxygen requirement (Yes, No)
- Region (US, ex-US)

Stratification discrepancies between the IXRS and the clinical database will be reviewed and assessed. The values recorded in the clinical database will be used for analyses in case there are discrepancies. Based on the assessment of stratification discrepancies, a sensitivity analysis of the primary endpoint may be performed.

The primary efficacy endpoint and the key  $\alpha$ -controlled secondary efficacy endpoint (see Section 6 for definition) will be evaluated in a stratified analysis based on the same 3 factors used for randomization, as specified in Section 6. In addition, observed imbalances between treatment groups in other baseline characteristics may be considered as covariates in sensitivity analyses of efficacy endpoints.

# 3.4. Examination of Participant Subgroups

The primary efficacy endpoint and the key  $\alpha$ -controlled secondary efficacy endpoint will be examined for the following participant subgroups:

- Kidney disease status (defined as: AKI, CKD and ESKD.)
- High-flow oxygen requirement at baseline (Yes, No)
- Region (US, ex-US)
- Participant's age ( $\geq 18 < 65, \geq 65 \text{ years}$ )
- Sex at birth: (a) male and (b) female
- Race: (a) Asian, (b) Black, (c) White, (d) Other
- Baseline risk factor (as applicable): Chronic lung disease (Yes, No), Hypertension (Yes, No), Cardiovascular or cerebrovascular disease (Yes, No), Diabetes mellitus (Yes, No), BMI (with categories: < 20, ≥ 20 < 30, ≥ 30 kg/m<sup>2</sup>), Immunocompromised state (Yes, No), Chronic liver disease (Yes, No), Current cancer (Yes, No)

In addition, the primary efficacy endpoint will be examined for duration of symptoms prior to first dose of study drug (<= 5 days vs >5 days) and baseline oxygen support status. Other subgroups may be considered based on imbalances between treatment groups observed in other baseline characteristics.

#### 3.5. Multiple Comparisons

To control the overall Type I error in the evaluation of the primary efficacy endpoint and the key secondary efficacy endpoint, the hypothesis testing will be performed in sequential order.

The primary efficacy endpoint will be tested first at the significance level of 0.05. If the primary efficacy endpoint null hypothesis is rejected, the key secondary efficacy endpoint will be tested at the 0.05 significance level; otherwise, the key secondary efficacy endpoint will not be tested.

All other endpoints may be tested using 2-sided tests at the 0.05 significance level without multiplicity adjustment as they are considered secondary CCI endpoints.

## 3.6. Missing Data and Outliers

## 3.6.1. Missing Data

In general, missing data will not be imputed unless methods for handling missing data are specified. Exceptions are presented in this document.

In this study, a missing pre-treatment laboratory result would be treated as normal (ie, no toxicity grade) for the laboratory abnormality summary.

For missing last dose date of study drug, imputation rules are described in Section 3.8.1. The handling of missing or incomplete dates for AE onset is described in Section 7.1.5.2, and for concomitant medications in Section 7.4.

Imputation rules for the secondary efficacy endpoints related to the 8-point ordinal scale score are described in Section 6.2.

#### **3.6.2. Outliers**

Outliers will be identified during the data management and data analysis process. No sensitivity analyses to evaluate the impact of outliers on efficacy or safety outcomes are planned. Unless specified otherwise, all data will be included in the analyses.

#### 3.7. Data Handling Conventions and Transformations

In general, age collected at Day 1 (in years) will be used for analyses and presented in listings. If age at Day 1 is not available for a participant, then age derived from date of birth and the Day 1 visit date will be used instead. If an enrolled participant was not dosed with any study drug, the randomization date will be used instead of the Day 1 visit date. For screen failures, the date the first informed consent was signed will be used for the age derivation. Age required for longitudinal and temporal calculations and analyses (e.g., estimates of creatinine clearance, age at date of AE) will be based on age derived from date of birth and the date of the measurement or event, unless otherwise specified.

The following conventions will be used for the imputation of date of birth when it is partially missing or not collected:

- If only year of birth is collected, then "01 July" will be imputed as the day and month of birth
- If year of birth is missing, then date of birth will not be imputed.

Laboratory data that are continuous in nature but are less than the lower LOQ or above the upper LOQ will be imputed as follows:

- A value that is 1 unit less than the LOQ will be used to calculate descriptive statistics if the datum is reported in the form of "< x" (where x is considered the LOQ). For example, if the values are reported as < 50 and < 5.0, values of 49 and 4.9, respectively, will be used to calculate summary statistics. An exception to this rule is any value reported as < 1 or < 0.1, etc. For values reported as < 1 or < 0.1, a value of 0.9 or 0.09, respectively, will be used to calculate summary statistics.
- A value that is 1 unit above the LOQ will be used to calculate descriptive statistics if the
  datum is reported in the form of "> x" (where x is considered the LOQ). Values with decimal
  points will follow the same logic as above.
- The LOQ will be used to calculate descriptive statistics if the datum is reported in the form of "\le x" or "\ge x" (where x is considered the LOQ).



Natural logarithm transformation will be used for analyzing concentrations. Concentration values that are BLQ will be presented as "BLQ" in the concentration data listing. Values that are BLQ will be treated as 0 at predose time points, and one-half the value of the LOQ at postdose time points for summary purposes.

The following conventions will be used for the presentation of summary and order statistics:

- If at least 1 participant has a concentration value of BLQ for the time point, the minimum value will be displayed as "BLQ."
- If more than 25% of the participants have a concentration data value of BLQ for a given time point, the minimum and Q1 values will be displayed as "BLQ."

- If more than 50% of the participants have a concentration data value of BLQ for a given time point, the minimum, Q1, and median values will be displayed as "BLQ."
- If more than 75% of the participants have a concentration data value of BLQ for a given time point, the minimum, Q1, median, and Q3 values will be displayed as "BLQ."
- If all participants have concentration data values of BLQ for a given time point, all order statistics (minimum, Q1, median, Q3, and maximum) will be displayed as "BLQ."

## 3.8. Analysis Visit Windows

## 3.8.1. Definition of Study Day

Study day will be calculated from the first dosing date of study drug and derived as follows:

- For assessment dates on or after the first dosing date: Assessment Date First Dosing Date + 1
- For assessment dates prior to the first dosing date: Assessment Date First Dosing Date

Therefore, Study Day 1 is the day of first dose of study drug administration.

Last Dose Date is defined as the maximum, nonmissing, nonzero dose end date of treatment recorded on the Study Drug Administration eCRF form with "Study Drug Permanently Withdrawn" box checked for participants who prematurely discontinued or completed study drug according to the Study Drug Completion eCRF.

Last dose date is not expected to be missing. However, if last dose date is missing, it will be imputed using the maximum of non-missing, non-zero dose, study drug start and stop dates.

Last Study Date is the latest of study drug start dates and end dates, the in-person or phone visit dates, the vital sign and the laboratory collection dates, including the Day 60 phone follow-up visit date. For participants who died during the study, the death date will be the Last Study Date. For participants who died after completing the study or after prematurely discontinuing the study, the death date will not be considered for the Last Study Date.

#### 3.8.2. Analysis Visit Windows

Participant visits might not occur on protocol-specified days. Therefore, for the purpose of analysis, observations will be assigned to analysis windows.

The analysis windows for chemistry (except for SCr), hematology and coagulation laboratory tests are provided in Table 3-1.

Table 3-1. Analysis Visit Windows for Chemistry (Except for SCr), Hematology, and Coagulation Laboratory Tests

| | | Visit Window Study Day | |
|---------------|-------------------|------------------------|--------------|
| Nominal Visit | Nominal Study Day | Lower Limit | Upper Limit |
| Baseline | 1 | (none) | 1 (Pre Dose) |
| Day 3 | 3 | 1 (Post Dose) | 3 |
| Day 5 | 5 | 4 | 6 |
| Day 8 | 8 | 7 | 10 |
| Day 12 | 12 | 11 | 14 |
| Day 16 | 16 | 15 | 18 |
| Day 20 | 20 | 19 | 22 |
| Day 24 | 24 | 23 | 26 |
| Day 29 | 29 | 27 | 44 |



The 8-point ordinal scale will be collected daily from Day 1 through Day 29 or discharge, whichever is earlier, as well as at the Day 29 and Day 60 phone follow-up. The analysis visit window will coincide with each study day up to Day 44 with 1 exception: a Day 1 postdose record will be mapped to Analysis Day 2 visit (the 8-point ordinal scale will be collected twice on Day 1: predose and the worst score on Day 1 post-dose). If any additional records are collected after Day 44, the analysis window is provided in Table 3-3.

Table 3-3. Analysis Visit Window for 8-Point Ordinal Scale Collected after Day 44

| | Nominal<br>Study Day | Visit Window Study Day | |
|---------------|----------------------|------------------------|-------------|
| Nominal Visit | | Lower Limit | Upper Limit |
| Day 60 | 60 | 45 | (none) |

Vital signs, and SCr will be collected daily from Day 1 through Day 29 or discharge, whichever is earlier, per protocol; therefore, the analysis visit window will coincide with each study day up to Day 29 with 1 exception: a Day 1 postdose record will be mapped to Analysis Day 2 visit.

# 3.8.3. Selection of Data in the Event of Multiple Records in an Analysis Visit Window

Depending on the statistical analysis method, single values may be required for each analysis window. For example, change from baseline by visit usually requires a single value, whereas a time-to-event analysis would use all data regardless of analysis window.

If multiple valid, nonmissing measurements exist in an analysis window, records will be chosen based on the following rules if a single value is needed:

- For baseline, the last nonmissing value on or prior to the first dosing date (and time,
  if available) of study drug will be selected, unless specified differently. If there are multiple
  records with the same time or no time recorded on the same day, the baseline value will be
  selected as follows:
  - For continuous data:
    - CCI
    - For other continuous data, the average of the measurements will be taken.
  - For categorical data:
    - For SARS-CoV-2 infection status, the highest severity (ie, a positive PCR result) will be selected.
    - For other categorical data, the lowest severity will be selected.

For the 8-point ordinal scale, only Screening and Day 1 predose values will be considered for baseline value selection.





In an analysis window (including baseline window), if both central lab and local lab results are available, then central lab results will be used for record selection instead of local lab results; local lab results will only be used for record selection if central lab results are missing.

## 3.9. Change from Protocol-Specified General Considerations

The multiplicity adjustment specified in the protocol Section 8.7 was changed because the interim analysis planned after 50% of participants completed the Day 29 assessment was not performed due to the stop of study enrollment prior to reaching 50% of planned enrollment. As there was no interim analysis, there was no alpha spent and the final analysis is planned at the 0.05 significance level (see Section 2.3).

#### 4. PARTICIPANT DISPOSITION

# 4.1. Participant Enrollment and Disposition

A table of key study dates will be provided, including first participant screened, first participant enrolled, last participant last visit for the primary endpoint, and last participant last visit.

The number and percentage of participants enrolled at each investigator site and country will be summarized by treatment group and overall. The denominator for this calculation will be the number of participants analyzed for that column.

A similar enrollment table will be provided by randomization stratum. The denominator for the percentage of participants in the stratum will be the total number of participants in the Safety Analysis Set. If there are discrepancies in the value used for stratification assignment between the IXRS and the clinical database, the value collected in the clinical database will be used for the summary. A listing of participants with discrepancies in the value used for stratification assignment between the IXRS and the clinical database at the time of data finalization will be provided.

A summary of participant disposition will be provided by treatment group and overall for all screened participants. This summary will include the number of participants screened, screen failure participants who were not randomized, participants who met all eligibility criteria but were not randomized, participants randomized, participants randomized but never treated, participants in the Safety Analysis Set, and Full Analysis Set (FAS).

In addition, the number and percentage of the participants in the following categories will be summarized:

- Completed study drug
- Did not complete study drug with reasons for premature discontinuation of study drug
- Completed study
- Did not complete study with reasons for premature discontinuation of study

The denominator for the percentages of participants in each category will be the number of participants in the Safety Analysis Set corresponding to that column.

No inferential statistics will be generated. A data listing of reasons for premature study drug/study discontinuation will be provided.

A summary of analysis sets will also be provided by treatment group and overall.

# 4.2. Extent of Study Drug Exposure

Number of doses received will be summarized by treatment group for the Safety Analysis Set.

#### 4.3. Protocol Deviations

A listing will be provided for all randomized participants who violated at least 1 inclusion or exclusion criterion. The listing will include the criteria not met.

Protocol deviations occurring after participants entered the study are documented during routine monitoring. The number and percentage of participants with important protocol deviations and the total number of important protocol deviations by deviation reason (eg, violation of select inclusion/exclusion criteria) will be summarized by treatment group for the FAS. A by-participant listing will be provided for those participants with important protocol deviations.

#### 5. BASELINE CHARACTERISTICS

# 5.1. Demographics and Baseline Characteristics

Participant demographic data (eg, sex, race, race category, ethnicity, age, and age group [< 18,  $\geq$  18 - < 65,  $\geq$  65 years]) and baseline characteristics (eg, body weight, height, body mass index [BMI] and BMI group [< 20,  $\geq$  20 - < 30,  $\geq$  30 kg/m^2]) will be summarized by treatment group and overall using descriptive statistics (n, mean, SD, median, Q1, Q3, minimum, and maximum) for continuous data and by the number and percentage of participants for categorical data. The summaries of demographic data and baseline characteristics will be provided for the Safety Analysis Set.

For categorical data, the Cochran-Mantel-Haenszel (CMH) test (ie, general association statistic for nominal data and row mean scores differ statistic for ordinal data) will be used to compare the 2 treatment groups. For continuous data, the 2-sided Wilcoxon rank sum test will be used to compare the 2 treatment groups.

Similar summaries will be produced for the following subgroups: kidney disease status (as defined in Section 3.4), high-flow oxygen requirement (Yes, No), and region (US vs. ex-US).

A by-participant demographic listing will be provided.

#### **5.2.** Other Baseline Characteristics

The following baseline disease characteristics will be summarized by treatment group and overall using descriptive statistics:

- Kidney disease status (as defined in Section 3.4)
- High-flow oxygen requirement (Yes, No)
- Region (US, ex-US)
- Clinical status (8-point ordinal scale)
- Oxygen support status
- RRT at baseline
- Duration of hospitalization prior to first dose of study drug
- Duration of symptoms prior to first dose of study drug (as a continuous variable, and a categorical variable with categories of <= 5 and > 5)
- Duration from SARS-CoV-2 positive result to first dose of study drug

- Alanine aminotransferase (ALT)
- Baseline risk factor (as defined in Section 3.4 except BMI)
- COVID-19 vaccine (See Appendix 2) status

For categorical data, the CMH test (ie, general association statistic for nominal data and row mean scores differ statistic for ordinal data) will be used to compare the 2 treatment groups. For continuous data, the 2-sided Wilcoxon rank sum test will be used to compare the 2 treatment groups.

Similar summaries will be produced for the following subgroups: kidney disease status (as defined in Section 3.4), high-flow oxygen requirement (Yes, No), and region (US vs. ex-US).

A by-participant listing will also be provided.

## 5.3. Medical History

General medical history data will be collected at screening. It will be coded using the current version of MedDRA.

A summary table will present the percentages of participants reporting each medical history preferred term, sorted first in alphabetical order by system organ class (SOC) and then by preferred term (PT) in descending order of total frequency within SOC. A listing of medical history will be provided.

A by-participant listing of kidney transplant history will also be provided.

#### 6. EFFICACY ANALYSES

# 6.1. Primary Efficacy Endpoint

## 6.1.1. Definition of the Primary Efficacy Endpoint

The primary endpoint is the composite of all-cause mortality or IMV from date of first dose through Day 29.

#### 6.1.2. Statistical Hypothesis for the Primary Efficacy Endpoint

**Null hypothesis**: There is no difference between treatment groups in the probability of all-cause mortality or IMV through Day 29.

**Alternative hypothesis**: The probability of all-cause mortality or IMV through Day 29 is different between treatment groups.

## 6.1.3. Primary Analysis of the Primary Efficacy Endpoint

The primary endpoint will be analyzed using a stratified log-rank test stratified by the randomization strata. P value and the proportion of all-cause mortality or IMV at Day 29 from Kaplan-Meier estimate will be provided.

The hazard ratio and 95% confidence interval (CI) will be estimated using a Cox model with stratification factors as covariates.

Participants with missing outcomes for the primary endpoint due to premature discontinuation of the study on or prior to Day 29 will be censored at the last study day.

Additionally, the difference in proportions of all-cause mortality or IMV at Day 29 between treatment groups and the 95% CI for the difference will be provided based on the stratum-adjusted Mantel-Haenszel (MH) proportion as described in {Koch 1989} in Appendix 2.

The FAS will be the primary analysis set for efficacy endpoint evaluation.

## 6.1.4. Secondary Analyses of the Primary Efficacy Endpoint

The primary endpoint will also be analyzed for each of the subgroups defined in Section 3.4.

Sensitivity analyses maybe conducted using the following alternative approaches for the primary endpoint.

• A CMH test including stratification factors as strata for the statistical comparison between treatment groups. If a participant prematurely discontinues from the study prior to Day 29 with no event before discontinuation or the IMV/death status is missing, the participant will be considered as with no IMV/death.

• In rare occasions, a participant may be unblinded to site for safety considerations (Gilead remains blinded). Data for such participants after site unblinding may be censored for a sensitivity evaluation.

The sensitivity analyses are for the purposes of evaluating the robustness of the estimates of the primary analysis.

## 6.2. Secondary Efficacy Endpoints

The key  $\alpha$ -controlled secondary endpoint is all-cause mortality through Day 29.

Other secondary endpoints include:

- Initiation of IMV through Day 29
- Time to recovery through Day 29
- Clinical status assessed by the 8-point ordinal scale at Day 15 and Day 29
- RRT-free days (among those without ESKD at baseline) through Day 29
- Proportion of participants with recovery through Day 29

Recovery is defined as achieving category 1, 2, or 3 on the 8-point ordinal scale score, for participants with a baseline score  $\geq 4$ .

## 6.2.1. Analysis of Secondary Efficacy Endpoints

The key  $\alpha$ -controlled secondary endpoint of all-cause mortality through Day 29 will be analyzed in a similar manner to the primary endpoint.

Initiation of IMV through Day 29 and time to recovery through Day 29 will also be analyzed in a similar manner to the primary endpoint except that a competing risk analysis approach will be used with death as the competing risk.

For analysis on time to recovery through Day 29, two sets of analyses will be conducted: (1) Time to recovery through Day 29, in which the first recovery without further worsening in the ordinal scale score (ie, a score of > 4) by Day 29 will be considered an event; (2) Time to recovery through Day 29, in which the first recovery (regardless of further worsening or not) will be considered an event.

The clinical status assessed by the 8-point ordinal scale at Day 15 and Day 29 will be analyzed using a proportional odds model including treatment as the independent variable. Two models will be explored; one with baseline score as a continuous covariate and one without baseline score as a covariate. The odds ratio and 95% CI will be provided. The percentage of participants in each category will be summarized by treatment group. The assumption of odds proportionality will be assessed using a score test and reported. Clinical status by study day and change from baseline up to Day 29 will also be summarized by treatment group.

For participants without ESKD at baseline, the number of RRT-free days will be calculated between date of first dose and Day 29. The number of RRT-free days will be calculated as the number of full days from Day 1 to Day 29 that the participant was alive and did not receive RRT. The number of RRT-free days will be summarized by treatment group, and compared between treatment groups using Wilcoxon rank sum test.

The proportion of participants with recovery through Day 29 will be summarized by treatment group, and compared between treatment groups using the CMH test stratified by randomization strata. Similar for time to recovery analysis, two sets of analyses will be conducted: (1) The proportion of participants with recovery through Day 29, in which recoveries without further worsening by Day 29 is considered; (2) The proportion of participants with recovery through Day 29, in which recoveries regardless of worsening status by Day 29 is considered.

The key  $\alpha$ -controlled secondary endpoint of all-cause mortality through Day 29 will also be analyzed for each of the subgroups defined in Section 3.4. Other secondary endpoints may also be analyzed for each of the stratification factor subgroups.

For time to event analysis of secondary endpoints, participants with missing outcomes due to premature discontinuation of the study on or prior to Day 29 will be censored at the date of last known status for that endpoint.

Clinical status assessed by the 8-point ordinal scale will be derived by combining the available death, hospital discharge alive and ordinal scale assessment reported by the site, where death supersedes discharge alive and discharge alive supersedes the ordinal scale score reported by the site.

Sites were instructed to report the worst ordinal scale category for each day. Therefore, the ordinal scale result on the day the participant was discharged alive does not necessarily reflect Not hospitalized. The definition of clinical status based on the 8-point ordinal scale is defined as follows:

- If a participant dies on or prior to Day 29, clinical status on the day of death and all subsequent days through Day 29 will be set as 8 (death)
- If a participant is discharged alive on or prior to Day 29, clinical status on the day of discharge alive will be set to 2 (not hospitalized, limitation on activities and/or requiring home oxygen), which is the worst score for a non-hospitalized participant
- If a participant is discharged alive and subsequently re-admitted on or prior to Day 29, and the 8-point ordinal score is not reported on the day of re-admission, the clinical status on the day of the re-admission will be imputed to 7 (hospitalized, on IMV or ECMO), which is the worst score for a hospitalized participant
- For other missing ordinal scores from Day 2 through Day 29, the clinical status will be imputed using the previous day's score (either reported score or imputed score as applicable)

The FAS will be the primary analysis set for the secondary efficacy endpoints.







# 6.4. Changes from Protocol-Specified Efficacy Analyses

The primary analysis specified in the protocol Section 8.2.2 and the final analysis will be combined into one final analysis due to early study closure with smaller than planned sample size.

#### 7. SAFETY ANALYSES

#### 7.1. Adverse Events and Deaths

## 7.1.1. Adverse Event Dictionary

Clinical and laboratory AEs will be coded using the current version of MedDRA. System organ class (SOC), high-level group term (HLGT), high-level term (HLT), preferred term (PT), and lower-level term (LLT) will be provided in the AE dataset.

#### 7.1.2. Adverse Event Severity

The severity of AEs will be graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 dated July 2017. For each episode, the highest grade attained should be reported as defined in the grading scale. The DAIDS scale is available at the following location:

https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf

Adverse events are graded by the investigator as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (life threatening) or Grade 5 (fatal) according to toxicity criteria specified in the document above. The severity grade of events for which the investigator did not record severity will be left as "missing" for data listings.

# 7.1.3. Relationship of Adverse Events to Study Drug

Related AEs are those for which the investigator selected "Related" on the AE CRF to the question of "Related to Study Treatment." Relatedness will always default to the investigator's choice, not that of the medical monitor. Events for which the investigator did not record relationship to study drug will be considered related to study drug for summary purposes. However, by-participant data listings will show the relationship as missing.

## 7.1.4. Serious Adverse Events

Serious adverse events (SAEs) will be identified and captured as SAEs if the AEs met the definitions of SAEs that were specified in the study protocol. SAEs captured and stored in the clinical database will be reconciled with the SAE database from the Gilead Global Patient Safety (GLPS) Department before data finalization.

## 7.1.5. Treatment-Emergent Adverse Events

#### 7.1.5.1. Definition of Treatment-Emergent Adverse Events

Treatment-emergent adverse events (TEAEs) are defined as 1 or both of the following:

- Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug
- Any AEs leading to premature discontinuation of study drug.

## 7.1.5.2. Incomplete Dates

If the onset date of the AE is incomplete and the AE stop date is not prior to the first dosing date of study drug, then the month and year (or year alone if month is not recorded) of onset determine whether an AE is treatment emergent. The event is considered treatment emergent if both of the following 2 criteria are met:

- The AE onset date is the same as or after the month and year (or year) of the first dosing date of study drug, and
- The AE onset date is the same as or before the month and year (or year) of the date corresponding to 30 days after the date of the last dose of study drug

An AE with completely missing onset and stop dates, or with the onset date missing and a stop date later than the first dosing date of study drug, will be considered treatment emergent. In addition, an AE with the onset date missing and incomplete stop date with the same or later month and year (or year alone if month is not recorded) as the first dosing date of study drug will be considered treatment emergent.

#### 7.1.6. Summaries of Adverse Events and Deaths

TEAEs will be summarized based on the Safety Analysis Set.

A brief, high-level summary of the number and percentage of participants who experienced at least 1 TEAE in the categories described below will be provided by treatment group. Treatment-emergent deaths observed in the study will also be included in this summary.

Treatment-emergent death refers to deaths that occurred between the first dose date and the last dose date plus 30 days (inclusive).

The number and percentage of participants who experienced at least 1 TEAE will be provided and summarized by SOC, High level term (HLT), PT, and treatment group.

For other AEs described below, summaries will be provided by SOC, PT, and treatment group:

- TEAEs with Grade 3 or higher
- TE study drug-related AEs
- TE study drug-related AEs with Grade 3 or higher
- TE SAEs
- TE study drug-related SAEs
- AEs leading to premature discontinuation of study drug

Multiple events will be counted only once per participant in each summary. Adverse events will be summarized and listed first in alphabetic order of SOC (and HLT within each SOC if applicable), and then by PT in descending order of total frequency within each SOC. For summaries by severity grade, the most severe grade will be used for those AEs that occurred more than once in an individual participant during the study.

In addition to the above summary tables, all TEAEs, TEAEs with Grade 3 or higher, TE study drug-related AEs, TE study drug-related AEs with Grade 3 or higher, and TE SAEs will be summarized by PT only, in descending order of total frequency.

The above summary tables may also be provided for one or more of the following subgroups: kidney disease status (as defined in Section 3.4), high-flow oxygen requirement (Yes, No), and/or region (US, ex-US).

In addition, data listings will be provided for the following:

- All AEs
- All study drug-related AEs
- All AEs with severity of Grade 3 or higher
- All SAEs
- All study drug-related SAEs
- All Deaths
- AEs leading to premature discontinuation of study drug

Listing of renal and hepatic adverse events will be provided. Hypersensitivity including infusion-related reactions adverse events will also be summarized and listed (See Appendix 2).

## 7.2. Laboratory Evaluations

Laboratory data collected during the study will be analyzed and summarized using both quantitative and qualitative methods. Summaries of laboratory data will be provided for the Safety Analysis Set and will include data collected up to the last dose of study drug plus 30 days. The analysis will be based on values reported in conventional units. When values are below or above the LOQ, they will be listed as such, and the closest imputed value will be used for the purpose of calculating summary statistics as specified in Section 3.7.

Because RRT may significantly impact certain lab values such as SCr and BUN, a sensitivity analysis will be conducted, in which records and/or participants may be excluded from analysis as follows:

• SCr and BUN will only be analyzed for participants who are not on RRT at baseline. If RRT is used during the study, any records from RRT start to end + 3 days will be excluded from analysis.

RRT started within 3 days before first dose is considered RRT at baseline.

Anticoagulation medications can impact coagulation lab parameters, such as aPTT, PT, and INR. Sensitivity analysis will be conducted for coagulation lab parameters. Any coagulation lab records under the influence of these medications will be excluded from analysis. For anticoagulation medications in the Warfarin class, coagulation lab records with a date in between the start and 5 + the stop date of the medication will be excluded; for other anticoagulation medications, records with a date in between the start and 1 + the stop date of the medication will be excluded.

A by-participant listing for laboratory test results will be provided by participant ID number and visit in chronological order for hematology, coagulation, serum chemistry. CCI

Values falling outside of the relevant reference range and/or having a severity grade of 1 or higher on the DAIDS Grading Scale (see Section 7.2.2) will be flagged in the data listings, as appropriate.

## 7.2.1. Summaries of Numeric Laboratory Results

Descriptive statistics will be provided by treatment group for selected laboratory test specified in the study protocol as follows:

- Baseline values
- Values at each postbaseline analysis visit
- Change from baseline at each postbaseline analysis visit
- Percentage change from baseline to each postbaseline analysis visit (if specified)

A baseline laboratory value will be defined as the last nonmissing measurement obtained on or prior to the date/time of first dose of study drug. Change from baseline to a postbaseline visit will be defined as the visit value minus the baseline value. The mean, median, Q1, Q3, minimum, and maximum values will be displayed to the reported number of digits; SD values will be displayed to the reported number of digits plus 1. Baseline and change from baseline will be compared between the treatment groups using the 2-sided Wilcoxon rank sum test.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3.

In an analysis window (including baseline window), if both central lab and local lab results are available, then central lab results will be used instead of local lab results; local lab results will only be used if central lab results are missing.

#### 7.2.2. Graded Laboratory Values

The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Event, Version 2.1 (July 2017) (see Section 7.1.2) will be used for assigning toxicity grades (0 to 4) to laboratory results for analysis. Grade 0 includes all values that do not meet the criteria for an abnormality of at least Grade 1. For laboratory tests with criteria for both increased and decreased levels, analyses for each direction (i.e., increased, decreased) will be presented separately.

For baseline, if both central lab and local lab results are available, then central lab results will be used to determine baseline toxicity grade; local lab results will only be used if central lab results are missing. For postbaseline laboratory abnormalities, both central lab and local lab results will be used.

# 7.2.2.1. Treatment-Emergent Laboratory Abnormalities

Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of study drug plus 30 days. If the relevant baseline laboratory value is missing, any abnormality of at least Grade 1 observed within the time frame specified above will be considered treatment emergent.

## 7.2.2.2. Summaries of Laboratory Abnormalities

Laboratory data that are categorical will be summarized using the number and percentage of participants in the study with the given response at baseline and each scheduled postbaseline visit.

The following summaries (number and percentage of participants) for treatment-emergent laboratory abnormalities will be provided by lab test and treatment group; participants will be categorized according to the most severe postbaseline abnormality grade for a given lab test:

- Treatment-emergent laboratory abnormalities
- Treatment-emergent Grade 3 or 4 laboratory abnormalities

For all summaries of laboratory abnormalities, the denominator is the number of participants with nonmissing postbaseline values up to 30 days after last dosing date.

A by-participant listing of treatment-emergent Grade 3 or 4 laboratory abnormalities will be provided by participant ID number and visit in chronological order.

# 7.2.3. Liver-Related Laboratory Evaluations

Liver-related abnormalities after initial study drug dosing will be examined and summarized using the number and percentage of participants who were reported to have the following laboratory test values for postbaseline measurements:

- Alanine aminotransferase (ALT): (a) > 3 × ULN, (b) > 5 × ULN, (c) > 10 × ULN,
   (d) > 20 × ULN
- Aspartate aminotransferase (AST): (a) > 3 × ULN, (b) > 5 × ULN, (c) > 10 × ULN,
   (d) > 20 × ULN
- ALT or AST: (a)  $> 3 \times ULN$ , (b)  $> 5 \times ULN$ , (c)  $> 10 \times ULN$ , (d)  $> 20 \times ULN$
- Total bilirubin: (a)  $> 1 \times ULN$ , (b)  $> 2 \times ULN$
- Alkaline phosphatase (ALP)  $> 1.5 \times ULN$
- ALT or AST  $> 3 \times$  ULN and total bilirubin: (a)  $> 1.5 \times$  ULN, (b)  $> 2 \times$  ULN
- ALT or AST  $> 3 \times ULN$  and total bilirubin  $> 2 \times ULN$  and ALP  $< 2 \times ULN$

For individual laboratory tests, participants will be counted once based on the most severe postbaseline value. For both the composite endpoint of ALT or AST and total bilirubin, and the composite endpoint of ALT or AST, total bilirubin, and ALP, participants will be counted once when the criteria are met at the same postbaseline visit date. The denominator is the number of participants in the Safety Analysis Set with nonmissing postbaseline value of the tests in evaluation at the same postbaseline visit date.

Listings of liver-related laboratory tests will be provided.

## 7.3. Vital Signs and Respiratory Status

Descriptive statistics will be provided by treatment group for vital signs (including pulse rate, respiratory rate and blood pressure) as follows:

- Baseline value
- Values at each postbaseline visit
- Change from baseline at each postbaseline visit

A baseline value will be defined as the last available value collected on or prior to the date/time of first dose of study drug. Change from baseline to a postbaseline visit will be defined as the postbaseline value minus the baseline value.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3. No formal statistical testing is planned.

A by-participant listing of vital signs (including pulse rate, temperature, blood pressure, height, weight, and respiratory rate) and respiratory status (including SpO<sub>2</sub>) will be provided by participant ID number and visit in chronological order.

#### 7.4. Concomitant Medications

Medications collected at screening and during the study will be coded using the current version of the World Health Organization (WHO) Drug dictionary.

Concomitant medications are defined as medications taken while a participant took study drug. Use of concomitant medications will be summarized by preferred name using the number and percentage of participants for each treatment group. A participant reporting the same medication more than once will be counted only once when calculating the number and percentage of participants who received that medication. The summary will be ordered by preferred name in descending overall frequency. For drugs with the same frequency, sorting will be done alphabetically.

For the purposes of analysis, any medications with a start date prior to or on the first dosing date of study drug and continued to be taken after the first dosing date, or started after the first dosing date but prior to or on the last dosing date of study drug will be considered concomitant medications. Medications started and stopped on the same day as the first dosing date or the last dosing date of study drug will also be considered concomitant. Medications with a stop date prior to the date of first dosing date of study drug or a start date after the last dosing date of study drug will be excluded from the concomitant medication summary. If a partial stop date is entered, any medication with the month and year (if day is missing) or year (if day and month are missing) prior to the date of first study drug administration will be excluded from the concomitant medication summary. If a partial start date is entered, any medication with the month and year (if day is missing) or year (if day and month are missing) after the study drug stop date will be excluded from the concomitant medication summary. Medications with completely missing start and stop dates will be included in the concomitant medication summary, unless otherwise specified. Summaries will be based on the Safety Analysis Set. No formal statistical testing is planned.

#### 7.5. Other Safety Measures

Renal replacement therapy during the study will be listed.

A data listing will be provided for participants experiencing pregnancy during the study.

# 7.6. Changes from Protocol-Specified Safety Analyses

There are no deviations from the protocol-specified safety analyses.




# 9. REFERENCES

Koch GG, Carr GJ, Amara IA, Stokes ME, Uryniak TJ. Categorical Data Analysis. Chapter 13 in Berry, D.A. (ed.). Statistical Methodology in the Pharmaceutical Sciences. New York: Marcel Dekker, Inc., 1989:pp. 414-21.

# 10. SOFTWARE

SAS® Software Version 9.4. SAS Institute Inc., Cary, NC, USA.

# 11. SAP REVISION

| Revision Date<br>(DD MMM YYYY) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|

# 12. APPENDICES

Appendix 1. Study Procedures Table
Appendix 2. Programming Specifications

# Appendix 1. Study Procedures Table

| | Screening | Baseline/<br>Day 1 | Day 2 | Day 3 | Day<br>4 | Day 5 | Day<br>6 | Day<br>7 | Day<br>8 | Day 9, 10, 11 | Day<br>12 | Day<br>13 | Day<br>14 | Day<br>15 | Day<br>16 | Day<br>17,<br>18,<br>19 | Day<br>20 | Day<br>21 | Day 22, 23 | Day<br>24 | Day<br>25,<br>26,<br>27,<br>28 | Day 29* | Day 29<br>and<br>Day 60<br>Phone<br>Follow-up<br>Visits<br>(+ 5 days) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Written Informed<br>Consent | X | | | | | | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion<br>Criteria | X | | | | | | | | | | | | | | | | | | | | | | |
| Focused Medical<br>History, including<br>SCr values <sup>a</sup> | X | | | | | | | | | | | | | | | | | | | | | | |
| Documentation of<br>SARS-CoV-2<br>Infection <sup>b</sup> | X | | | | | | | | | | | | | | | | | | | | | | |
| Complete Physical Examination | X | | | | | | | | | | | | | | | | | | | | | | |
| Height | X | | | | | | | | | | | | | | | | | | | | | | |
| Weight | X | | | | | | | | | | | | | | | | | | | | | | |
| Vital Signs <sup>c</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Respiratory Status <sup>d</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Invasive Mechanical Ventilation <sup>q</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Pulmonary<br>Radiographic<br>Imaging <sup>e</sup> | X | | | | | | | | | | | | | | | | | | | | | | |
| 8-Point Ordinal<br>Scale <sup>f</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pregnancy Test <sup>g</sup> | X | | | | | | | | | | | | | | | | | | | | | | |
| Chemistry <sup>h,r</sup> | X | X | | X | | X | | | X | | X | | | | X | | X | | | X | | X | |
| Hematology <sup>i,r</sup> | X | X | | X | | X | | | X | | X | | | | X | | X | | | X | | X | |
| Coagulation <sup>j,r</sup> | X | X | | X | | X | | | X | | X | | | | X | | X | | | X | | X | |
| Serum Creatininer,s | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |

Day 29

X

| | Screening | Baseline/<br>Day 1 | Day 2 | Day 3 | Day<br>4 | Day<br>5 | Day<br>6 | Day<br>7 | Day<br>8 | Day<br>9,<br>10, | Day<br>12 | Day<br>13 | Day<br>14 | Day<br>15 | Day<br>16 | Day<br>17,<br>18,<br>19 | Day<br>20 | Day<br>21 | Day 22, 23 | Day<br>24 | Day 25, 26, 27, 28 | Day 29* | and Day 60 Phone Follow-up Visits (+ 5 days) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Urinalysis <sup>t</sup> | X | | | | | | | | | | | | | | | | | | | | | | |
| RRT Assessmentk | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Virologic Testing <sup>l</sup> | | X | | X | | X | | X | | | | | X | | | | | X | | | | X | |
| CCI | | | | | | | | | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | | | | | | | | | |
| Investigational Drug<br>Dosing | | X | X | X | X | X | | | | | | | | | | | | | | | | | |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant<br>Medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Mortality | | | | | | | | | | | | | | | | | | | | | | | X |

- \* All assessments to be completed through Day 29, or until discharge, whichever is earlier. If participant is discharged prior to Day 29, a phone follow-up is to be completed at Day 29 and Day 60.
- a Focused medical history will include date of first symptoms, overall symptoms, exposure source, demographics, baseline characteristics, concomitant medications, kidney or other transplant history, and allergies. If available, up to 3 SCr values prior to COVID-19 illness (eg, within the previous 6 months) should be provided. Document COVID-19 vaccine status. (Note: It should be documented whether participant is fully or partially vaccinated, including any booster[s] received, if applicable.)
- b Positive as determined by PCR via 1 validated assay at a local laboratory, if not performed within the last 4 calendar days.
- $c \qquad \text{Includes heart rate, temperature, and blood pressure.} \\$

Hospital Readmission

Rate

- d Respiratory status includes respiratory rate and oxygenation: see protocol Sections 6.2.1, 6.2.2, and 6.4.
- e Pulmonary radiographic imaging may be performed within 72 hours, if not already available and if needed to satisfy eligibility criteria.

- f Ordinal scale to be performed twice on Day 1: prior to randomization (for baseline predose score) and the worst score on Day 1.
- g Serum pregnancy test will only be done for women of childbearing potential. Women < 54 years of age with amenorrhea of ≥ 12 months may also be considered postmenopausal if their follicle stimulating hormone (FSH) level is in the postmenopausal range > 40 IU/L and they are not using hormonal contraception or hormonal replacement therapy. Results from within 48 hours prior to screening are acceptable.
- h Chemistry: alkaline phosphatase, AST, ALT, total bilirubin, total protein, albumin, lactate dehydrogenase, creatine phosphokinase, bicarbonate, blood urea nitrogen, calcium, chloride, creatinine, glucose, lipase, magnesium, phosphorus, potassium, sodium, uric acid. Results from within 48 hours prior to screening are acceptable.
- i Hematology: complete blood count with differential, hemoglobin and/or hematocrit, platelets. Results from within 48 hours prior to screening are acceptable.
- j Coagulation performed by central lab: international normalized ratio, prothrombin time, activated partial thromboplastin time, D-dimer, fibrinogen. Results from within 48 hours prior to screening are acceptable.
- k RRT will be measured at screening through Day 29 or until discharge from inpatient hospitalization, as well as at the Day 60 phone follow-up.
- Nasopharyngeal swab collection for virologic (SARS-CoV-2) testing for participants on Days 1, 3, 5, 7, 14, 21, and 29 or until discharge, whichever is earlier.
- If on invasive mechanical ventilation at screening, participant should be excluded from the study.
- r For participants on intermittent RRT, laboratory safety assessments should be drawn before dialysis on the day of dialysis.
- s Refer to protocol Inclusion Criterion #5 to determine the need for a confirmatory SCr evaluation.
- t Participants who are oliguric are not required to provide a urine sample.

# **Appendix 2. Programming Specifications**

1) If the age from the Day 1 eCRF is not available, age will be calculated as follows:

Only year is provided for the date of birth (DOB). Use July 1 for the month and day.

- a) AGE (years) is calculated from the number of days between the DOB and Study Day 1,
- b) Use the SAS INTCK function to determine the number of "1st-of-month days" (eg, January 1st, February 1st, March 1st) between DOB and Day 1 (inclusive),
- c) Divide the result in (b) by 12,

AGE =the integer of the result in (c),

Age for laboratory test reference range will be based on the age at the sample collection date

- 2) All screened participants refer to all participants who are screened (ie, with non-missing screening date) and have a screening number. For summaries the same participant is counted only once.
- 3) Screen failure participants are the participants who were screened and answered "No" for any inclusion criteria or "Yes" for any exclusion criteria regardless of which version of protocol the participant was consent to.
- 4) Participants in the randomized analysis set are defined as participants randomized into the study. IXRSRAND is the source to determine whether the participant is randomized (ie, participant with non-missing RGMNDTN in the IXRSRAND dataset), and confirmed by the eCRF ENROLL dataset (ie, ENROLLYN = "Yes" in ENROLL dataset).
- 5) Randomized treatment (ie, TRT01P in ADSL) is derived from IXRSRAND, while actual treatment received (ie, TRT01A in ADSL) is assigned as the randomized treatment if participant took at least 1 dose of study drug and assigned as blank if the participant was never dosed.
- 6) In the disposition table, the reasons for premature discontinuation are displayed in the order as they appear on the eCRF.
- 7) Body mass index (BMI)

BMI will be calculated only at baseline as follows:

-- BMI = (weight [kg]) / (height [meters]<sup>2</sup>)

Baseline height and weight will be used for this calculation if available

#### 8) TEAE

# **Events with Missing Onset Day and/or Month**

An event is considered treatment emergent if all of the following 3 criteria are met:

- i. The month and year (or year) of onset date is the same as or after the month and year (or year) of the first dose of study drug, and
- ii. The month and year (or year) of the onset date is the same as or before the month and year (or year) of the 30th day after the date of the last dose of study drug, and
- iii. End date is as follows:

The (complete) end date is on or after the first dose date, or

The month and year (or year) of end date is the same or after the month and year (or year) of the first dose of study drug, or

End date is completely missing

# **Events with Completely Missing Onset Date**

An AE with a completely missing onset date is defined as TEAE if end date meets any of the 3 criteria specified above.

#### 9) Baseline risk factor

Selected medical history will be summarized as baseline risk factor and be included as subgroups in analysis. The risk factor of "current cancer" for a participant is defined as a medical history of one of these diseases:

- At least 1 ongoing medical history record with MedDRA PT (mh.MDRPT) in the following selected PT listing for the corresponding disease with start date on or prior to the first dose date;
- At least 1 ongoing AE record with MedDRA PT (ae.MDRPT) in the following selected PT listing for the corresponding disease with start date on or prior to the first dose date.

Other risk factors for a participant is defined as a medical history of one of these diseases:

- At least 1 medical history record with MedDRA PT (mh.MDRPT) in the following selected PT listing for the corresponding disease with start date on or prior to the first dose date;
- At least 1 AE record with MedDRA PT (ae.MDRPT) in the following selected PT listing for the corresponding disease with start date on or prior to the first dose date. If the start date is incomplete but the month and year (or year alone) of the start date is the same as or before the month and year (or year alone) of the first dosing date of study drug, the event will be included. If the start date is completely missing, the event will be included.

If the ongoing status is missing for an event:

- If the end date is completely missing and start date is the same as or before the first dosing date of the study drug, the event will be included;
- If the end date is completely missing and start date is after the first dosing date of the study drug, the event will not be included;
- If the end date is incomplete but the month and year (or year alone) of the end date is the same as or after the month and year (or year alone) of the first dosing date of study drug, the event will be included;
- If the end date is incomplete but the month and year (or year alone) of the end date is before the month and year (or year alone) of the first dosing date of study drug, the event will not be included.

A variable for each of the risk factors will be added to raw Medical History and Adverse Events datasets. A medical history or an AE record will be flagged for a risk factor if its MedDRA PT is included in the prespecified PT list for the corresponding disease of interest, which includes all PTs from the narrow or broad search of the following SMQs under MedDRA 25.0 provided by

| 0'1 1 OT DO | 1 | 1 . | O:1 1 | 1. 1 | • . |
|-------------------|--------------|-------|-----------|----------|------------|
| ( -1 lood ( -1 DV | and reviewed | hrr 1 | ( -11004 | madiant | monitora |
| CHIEAG CH P.S | and reviewed | 111/ | t tileaci | THECHCAL | HIIOHHIOIS |

| Disease of Interest | SMQ or MedDRA HLT Source |
|---|---|
| Chronic lung disease | HLT of bronchospasm and obstruction |
| Hypertension | Hypertension (SMQ) |
| Cardiovascular or cerebrovascular disease | Ischaemic central nervous system vascular conditions (SMQ); Myocardial infarction (SMQ); |
| | Other ischaemic heart disease (SMQ) |
| Diabetes mellitus | Hyperglycaemia/new onset diabetes Mellitus (SMQ) |
| Immunocompromised state | HLGT for "Immunodeficiency syndromes" |
| Chronic liver disease | search name "Chronic liver disease excluding transient_acute events and nonspecific signs_symptoms" |
| Current cancer | Malignancies (SMQ) |

10) Details on SCr and BUN record exclusion for sensitivity analysis

SCr and BUN will only be analyzed for participants who are not on RRT at baseline.

#### RRT at baseline:

RRT started within 3 days of first dose is considered RRT at baseline. An RRT record with an end date prior to the first dose date - 3 days (or 72 hours if time available) or a start date/time after the first dose date/time will not be considered a baseline RRT record; otherwise, the record will be considered baseline.

# SCr/BUN record exclusion (for participants who are not on RRT at baseline):

Any SCr/BUN records from an RRT start to end + 3 days will be excluded from analysis.

If both date and time are collected for RRT and labs, only date will be used, with 1 exception below:

If an SCr/BUN record is collected on the first dose date and prior to first dose time, and the participant's first RRT starts on the first dose date but after first dose time, then this lab record will not be excluded.

#### RRT date:

A missing end date of a hemodialysis record will be imputed using the hemodialysis start date.

If an end date is missing for a CVVH record:

- If this record is followed by another RRT (CVVH or hemodialysis) record, then the end date of this CVVH record will be imputed as the start date of the subsequent RRT record;
- If this record is the last available or the only RRT record for a participant:
  - If the participant died after the start of this CVVH record, then the end date of this CVVH record will be imputed as the death date;
  - Otherwise, the end date of this CVVH record will not be imputed, and all the SCr and BUN records after the start date of this CVVH record will be excluded from analysis.

#### 11) Details on coagulation lab record exclusion for sensitivity analysis

Any coagulation lab records under the influence of anticoagulation medications will be excluded from analysis. For coagulation lab record exclusion, the start/end date of anticoagulation medications will be used. An anticoagulation medication may be taken chronically prior to and/or during the study.

#### Anticoagulation medication date:

If a medication end date is missing, the medication will be considered as "ongoing", and all coagulation lab records after the medication start date will be excluded from analysis.

If a medication start date is missing, all coagulation lab records will be considered after the medication start date.

For a partial medication end date:

• If only date is missing, then the date will be imputed as the last date of the month;

• If both month and date is missing, then the month and date will be imputed as December 31st of the year.

For a partial medication start date:

- If only date is missing, then the date will be imputed as the first date of the month;
- If both month and date is missing, then the month and date will be imputed as January 1st of the year.
- 12) Treatment difference in percentages not adjusted by stratum

The percentage difference between two treatment groups and its 95% CIs are calculated based on the unconditional exact method using 2 inverted 1-sided tests in SAS v9.3 or above.

The following SAS code will be used to compute cell counts and p-values.

```
data example;
input grp trt $ outcome $ count;
datalines;
     Treat-A
                 2-Fail
                           X
1
     Treat-A
                 1-Succ
                          XXX
1
     Treat-B
                2-Fail
                          X
1
     Treat-B
                1-Succ
                          XXX
run:
proc freq data = example;
table trt*outcome /riskdiff(CL=(exact)) alpha=0.05;
weight count; exact RISKDIFF(METHOD=SCORE);
output out=ciexact(keep= RDIF1 XL RDIF1 XU RDIF1 RSK11 __ RSK21) riskdiff;
run;
data final(keep=A1 B1 Estimate LowerCL UpperCL ocharc1);
set ciexact;
label Estimate ="Percentage Difference"
LowerCL = "95% Lower Confidence Limit"
UpperCL = "95% Upper Confidence Limit"
A1 = "Percentage of Success in Treat-A"
B1 = "Percentage of Success in Treat-B";
Estimate=100* RDIF1;
LowerCL = 100*XL RDIF1;
UpperCL = 100*XU RDIF1;
A1 = 100* RSK11;
B1 = 100* RSK21 ;
ocharc1 = right(compress(put(Estimate, 8.1)) || '% (' || compress(put(LowerCL, 8.1)) || '%
to ' || compress(put(UpperCL, 8.1)) || '%)');
run;
```

# 13) Difference in proportions between treatment groups adjusted by stratum

The 95% confidence interval for difference in between treatment groups will be calculated based on the stratum-adjusted Mantel-Haenszel (MH) proportion as described as follows {Koch 1989}, where the stratification factors include ESKD (Yes, No), High-flow oxygen requirement (Yes, No), and region (US, ex-US):

$$P_1 - P_2 \pm Z_{(1-\alpha/2)} * SE(P_1 - P_2),$$

where

- $(P_1 P_2) = \frac{\sum w_h d_h}{\sum w_h}$ , is the stratum-adjusted MH proportion difference, where  $d_h = p_{1h} p_{2h}$  is the difference in the proportions of Treatment Groups 1 and 2 in stratum h.
- $W_h = \frac{n_{1h}n_{2h}}{n_{1h} + n_{2h}}$ , is the weight based on the harmonic mean of sample size per treatment group for each stratum where  $n_{1h}$  and  $n_{2h}$  are the sample sizes of the Treatment Groups 1 and 2 in stratum h.

• SE(P<sub>1</sub>-P<sub>2</sub>) = 
$$\sqrt{\frac{\sum \frac{p_{1h}^*(1-p_{1h}^*)}{n_{1h}-1} + \frac{p_{2h}^*(1-p_{2h}^*)}{n_{2h}-1}}{(\sum w_h)^2}}$$
, where  $p_{1h}^* = \frac{m_{1h}+0.5}{n_{1h}+1}$  and  $p_{2h}^* = \frac{m_{2h}+0.5}{n_{2h}+1}$ .  $m_{1h}$  and  $m_{2h}$  are the number of participants with event interest at Day 29 in Treatment Groups 1 and 2 in stratum  $h$ .

- $\alpha = 0.05$  for this study
- $Z_{(1-\alpha/2)} = Z_{0.975} = 1.96$  is the 97.5<sup>th</sup> percentile of the normal distribution

Note that if the computed lower confidence bound is less than -1, the lower bound is defined as -1. If the computed upper confidence bound is greater than 1, the upper bound is defined as 1.

To facilitate SAS macro use, a single stratum variable could be defined as:

| ESKD requiring chronic dialysis | High-flow oxygen requirement | Region | Stratum |
|---|---|---|---|
| Yes | No | US | 1 |
| Yes | No | ex-US | 2 |
| Yes | Yes | US | 3 |
| Yes | Yes | ex-US | 4 |
| No | No | US | 5 |
| No | No | ex-US | 6 |
| No | Yes | US | 7 |
| No | Yes | ex-US | 8 |

# 14) Clarification for SE(P1-P2) Calculation in 13).

- if n1h or n2h > 1 the denominator n1h 1 or n2h 1 was calculated as indicated in the formula:
- if n1h or n2h =1, the corresponding n1h or n2h will be adjusted to 2, then corresponding denominator [(n1h 1) or (n2h 1)] is 1;
- if n1h or n2h = 0, then the corresponding stratum will be ignored, will not be included in the calculation, thus the proportion difference and 95% CI are still calculable.

#### 15) Kidney disease status definition

Kidney disease data at baseline are collected in this study, including: history of CKD and ongoing AKI from the Medical History CRF form, ESKD status at Screening from the ENROLLMENT CRF form, and renal transplant history from the Transplant History CRF form.

Expected data patterns are as follows (renal transplant history can be present or absent for any of these combinations):

| | Ongoing AKI<br>(from MH CRF<br>question) | History of CKD<br>(from MH CRF<br>question) | ESKD status at Screening<br>(from ENROLLMENT<br>CRF) | Kidney Disease<br>Status |
|---|---|---|---|---|
| 1 | Yes | Any | No | AKI |
| 2 | No | Yes | No | CKD |
| 3 | Any | Any | Yes | ESKD |

Kidney disease status is defined as:

- AKI: the 1<sup>st</sup> row of the above table, ie, ongoing AKI with or without history of CKD
- CKD: the 2<sup>nd</sup> row of the above table, ie, history of CKD without ongoing AKI
- ESKD: the 3<sup>rd</sup> row of the above table.
- 16) For demographics tables, "Not Permitted" will be excluded from percentage for detailed race categories summary (ie, race categories collected on eCRF). For combined Race Category (e.g. Asian, White, Black, Other), "Not Permitted" is included in "Other" and "Other" will be included in the count of percentage.
- 17) For calculation of peak serum creatinine (SCr) through Day 29 (among those without ESKD at baseline), (1) baseline records will not be included; (2) Day 1 postdose is included in the calculation; (3) for multiple records within one day, the observed record with max SCr will be selected; (4) For multiple days has the same highest value, the earliest will be picked.

#### 18) Death date imputation

For a partial death date where the year and month are available but the date is missing, the following imputation will be performed:

- If the latest clinical date (ie, the latest of study drug start dates and end dates, the in-person or phone visit dates, the vital sign and the laboratory collection dates, including the Day 60 phone follow-up visit date) falls into the same year/month of death, then this latest clinical date will be used to impute the date of death;
- If the latest clinical date falls into the same year, but a prior month of death, then the 1<sup>st</sup> of the month of death will be the imputed date of death;
- If the latest clinical date falls into a prior year of death, then the 1<sup>st</sup> of the month of death will be the imputed date of death.
- 19) The precision in reporting numerical values should be as follows:

Raw measurements will be reported the same as the data captured electronically or on the eCRF.

Standard deviation and standard error will be reported to one more significant decimal place than the raw measurement.

Mean, median, minimum, Q1, Q3, maximum, 95% CIs will be reported to the same number of decimal places of the raw measurements.

If records for the same lab use different decimal places, the decimal place with majority records would be used.

Exceptions may be considered.

# 20) Graded Laboratory Abnormalities Summary

The following labels will be used for laboratory abnormalities and Grade 3 or 4 laboratory abnormalities summary tables and listings:

| Battery | Lab Test Label Used in<br>I-labtox Listing | Toxicity<br>Direction | Lab Test Label Used in t-labtox Table |
|---|---|---|---|
| | Hemoglobin | Decrease | Hemoglobin (Decreased) |
| | Lymphocytes | Decrease | Lymphocytes (Decreased) |
| Hematology | Neutrophils | Decrease | Neutrophils (Decreased) |
| | Platelets | Decrease | Platelets (Decreased) |
| | WBC | Decrease | WBC (Decreased) |
| | Albumin | Decrease | Albumin (Decreased) |
| | Alkaline Phosphatase | Increase | Alkaline Phosphatase (Increased) |
| | ALT | Increase | ALT (Increased) |
| | AST | Increase | AST (Increased) |
| | Bicarbonate | Decrease | Bicarbonate (Decreased) |
| | Corrected Calcium | Increase | Corrected Calcium (Hypercalcemia) |
| | Corrected Calcium | Decrease | Corrected Calcium (Hypocalcemia) |
| | Creatine Kinase (CK) | Increase | Creatine Kinase (Increased) |
| | Creatinine | Increase | Creatinine (Increased) |
| | Lipase | Increase | Lipase (Increased) |
| | Magnesium | Decrease | Magnesium (Hypomagnesemia) |
| Chemistry | Phosphate | Decrease | Phosphate (Hypophosphatemia) |
| | Serum Glucose | Increase | Serum Glucose (Hyperglycemia) |
| | Serum Glucose | Decrease | Serum Glucose (Hypoglycemia) |
| | Serum Potassium | Increase | Serum Potassium (Hyperkalemia) |
| | Serum Potassium | Decrease | Serum Potassium (Hypokalemia) |
| | Serum Sodium | Increase | Serum Sodium (Hypernatremia) |
| | Serum Sodium | Decrease | Serum Sodium (Hyponatremia) |
| | Total Bilirubin | Increase | Total Bilirubin (Hyperbilirubinemia) |
| | Uric Acid | Increase | Uric Acid (Hyperuricemia) |
| | Prothrombin Intl.<br>Normalized Ratio (INR) | Increase | Prothrombin Intl. Normalized Ratio (Increased) |
| Coagulation | Prothrombin Time (PT) | Increase | Prothrombin Time (Increased) |
| Coagulation | Activated partial thromboplastin time (aPTT) | Increase | Activated partial thromboplastin time (Increased) |

21) SAS codes for the treatment comparison for demographics and baseline characteristics tables.

CMH test for nominal variable (Y), the p-value from the general association test should be used for nominal variables:

```
proc freq;
tables trt * Y /cmh; /*general association test*/
run;
```

CMH test for ordinal variable (Y), the p-value from the row mean score test should be used for ordinal variables:

```
proc freq;
tables trt * Y / cmh2 ; /*row mean score test*/
run;
```

Wilcoxon rank sum test for continuous variable (Y), the p-value from the normal approximation two-sided test should be used for continuous variables:

```
proc nparlway wilcoxon;
class trt;
var Y;
run;
```

# 22) Proportional Odds

A proportional odds model including treatment as the independent variable and baseline score as a continuous covariate to compare the treatment groups:

```
proc logistic;
```

```
class trt/ param=ref order=data;
model outcome(descending)= trt baseline;
run;
```

A proportional odds model including treatment as the independent variable to compare the treatment groups (without covariate):

# proc logistic;

```
class trt/ param=ref order=data;
model outcome(descending)= trt;
run;
```

where outcome is the ordinal scale response at Day 15 and Day 29.

#### 23) Cox model:

a) with stratification factors as covariates

```
proc phreg;
class trt strat1 strat2 strat3;
model aval*cnsr(1) = trt strat1 strat2 strat3 /risklimits = wald;
ods output ParameterEstimates=Est1 ModelANOVA = pvout1;
run;
b) with no stratification factors as covariates
proc phreg;
class trt;
model aval*cnsr(1) = trt /risklimits = wald;
ods output ParameterEstimates=Est1 ModelANOVA = pvout1;
run;
```

# 24) log-rank test

Log-rank test between treatment groups:

```
proc lifetest;
time aval*cnsr(1);
strata trt;
run;
```

The binary indicator variable (cnsr) with a value of 0 indicates the time to the event of interest is complete or 1 indicates the time to the event is censored.

#### 25) Stratified log-rank test

Log-rank test between treatment groups:

```
proc lifetest;
time aval*cnsr(1);
strata strat1 strat2 strat3/group=trt;
run;
```

The binary indicator variable (cnsr) with a value of 0 indicates the time to the event of interest is complete or 1 indicates the time to the event is censored.

# 26) Competing risk analysis

The following SAS code will be used to generate the cause-specific hazard ratio and 95% confidence intervals for the competing risk analysis:

```
proc phreg;
class trt strat1 strat2 strat3;
model aval* cnsr (1, 2) = trt strat1 strat2 strat3 / rl;
hazardratio "Cause-specific hazard" trt;
run;
```

where cnsr = 0 if the participant had the event; cnsr = 2 if the participant died prior to having the event, and cnsr = 1 if the participant did not have the event and did not die.

SAS codes to obtain a cumulative incidence function plot and dataset for further processing for time to first event table:

```
proc lifetest outcif=outcif plots=cif;
strata trt;
time aval* cnsr (1) / failcode = 0;*Note: this produces data for the event of interest only;
run;
```

SAS code to obtain support tables:

```
proc univariate;
by trt cnsr;
var aval;
output pctlpre=P_ min=min max=max pctlpts= 10, 25, 50, 75, 90;
run;
```

27) SAS code for stratified 2-sided Wilcoxon Rank sum test (stratified on baseline result)

```
proc freq;
  table base*trt*aval/cmh2 scores=modridit;
run;
```

where BASE is the baseline value.

# 28) SAS code for ANCOVA:

```
ods output ParameterEstimates=out1 LSMeans=out2 LSMeanCL=out3 LSMeanDiffCL=out4;

proc glm data=dat1 plots=none;
class trt;
model DAVG = trt base / solution;
lsmeans trt / stderr cl pdiff;
run;
ods output close; quit;
```

29) SAS code for CMH test and estimates with stratification factors adjustment:

```
proc freq data=dat1;
  tables strat1*strat2*strat3*trt*Y/ list cmh;
ods output cmh=cmhpval CommonRelRisks=risk;
run;
```

- 30) Renal and hepatic adverse events include preferred terms from search term list 'Acute Renal Failure (SMQ)' and search term list 'Acute and non-infectious liver events' MedDRA 25.0.
- 31) Vital signs, and SCr collected after Day 29, PCR collected after day 44 will be assigned to "Post Day 29".

#### CC

- 33) For coagulation laboratory tests, both local and Covance lab records are collected in the data. In a visit where both Covance and local lab records are collected, Covance records will be picked over local lab records.
- 34) Reference ranges are based on Covance laboratory reference ranges.
- 35) COVID-19 medications include the following drugs:

| Drug name |
|--------------------------|
| Chloroquine |
| Hydroxychloroquine |
| Lopinavir/ritonavir |
| Ribavirin |
| Remdesivir |
| Bamlanivimab/ etesevimab |
| Casirivimab/Imdevimab |
| Molnupiravir |
| Monoclonal antibodies |
| Convalescent plasma |
| Sotrovimab |
| Nirmatrelvir |
| Paxlovid |
| Regdanivimab |
| Tixagevimab/cilgavimab |

# with preferred term codes (WHODrug BMAR2022):

| Prohibited PREF<br>Codes | Prohibited PREF<br>Codes | Prohibited PREF<br>Codes | Prohibited PREF<br>Codes | Prohibited PREF<br>Codes |
|---|---|---|---|---|
| 15665101001 | 14055301001 | 13983301001 | 13980301001 | 14248901001 |
| 15585401001 | 14068301001 | 14000901001 | 15847201001 | 08968801001 |
| 00001001001 | 15250901001 | 15337902001 | 08030701001 | 08342801001 |
| 00001002001 | 15379801001 | 15337901001 | 05699301001 | 15494501001 |
| 00001003001 | 15925301001 | 09304301001 | 14780501001 | 15646401001 |
| 00001004001 | 15701601001 | 15684201001 | 14780502001 | 15341201001 |
| 00001005001 | 15290701001 | 06356701001 | 15945601001 | 15633201001 |
| 00001006001 | 15251201001 | 14011101001 | 15395601001 | 15396501001 |
| 00001007001 | 15251601001 | 14033401001 | 14026001001 | 14048001001 |
| 00001008001 | 15416301001 | 15770001001 | 14056001001 | 01555211001 |
| 11198301001 | 15343501001 | 14182301001 | 14053601001 | 14057701001 |
| 11198302001 | 15665101001 | 14659001001 | 15356801001 | 14049401001 |
| 11282901001 | 15774801001 | 13408901001 | 14031801001 | 14010801001 |
| 11282902001 | 14037301001 | 15401601001 | 14492001001 | 01555207001 |
| 11617101001 | 14036401001 | 14816501001 | 14036601001 | 14548401001 |
| 11617102001 | 14052601001 | 14999701001 | 08032001001 | 14548402001 |
| 11724901001 | 14022401001 | 14033301001 | 01555212001 | 15400501001 |
| 11724902001 | 14148201001 | 14149501001 | 14164901001 | 15322701001 |
| 11725001001 | 13980701001 | 15350401001 | 13981101001 | 08969201001 |
| 11725002001 | 14022501001 | 15585401001 | 13983101001 | 08969202001 |
| 11725101001 | 15719902001 | 15710301001 | 15796001001 | 01402501001 |
| 11725102001 | 15719901001 | 15139201001 | 14691701001 | 01402503001 |
| 11725201001 | 13947301001 | 14183001001 | 14691702001 | 01402507001 |
| 11725202001 | 14152101001 | 14181701001 | 14057401001 | 01402502001 |
| 11725301001 | 13983001001 | 13999801001 | 15342201001 | 01402506001 |
| 11725302001 | 01555201001 | 15429101001 | 14039101001 | 01402504001 |
| 11725401001 | 01555202001 | 15616901001 | 14547901001 | 14055601001 |
| 11725402001 | 01555206001 | 13981201001 | 13978101001 | 14666201001 |
| 13117801001 | 01555205001 | 14004701001 | 08342601001 | 14346101001 |
| 13118301001 | 01555203001 | 14005201001 | 01555210001 | 07222101001 |
| 13118401001 | 12336402001 | 14031101001 | 14397901001 | 01555213001 |

| Prohibited PREF<br>Codes | Prohibited PREF<br>Codes | Prohibited PREF<br>Codes | Prohibited PREF<br>Codes | Prohibited PREF<br>Codes |
|---|---|---|---|---|
| 13183901001 | 14396302001 | 14001401001 | 14030401001 | 07244601001 |
| 13480201001 | 14396401001 | 07841501001 | 14585201001 | 06331801001 |
| 13480202001 | 14396501001 | 09304401001 | 14155601001 | 07209901001 |
| 14001301001 | 14396502001 | 09304402001 | 13979801001 | 15464401001 |
| 14001302001 | 14397801001 | 01445608001 | 15350501001 | 15429001001 |
| 14001303001 | 13975801001 | 12759302001 | 01445601001 | 01759101001 |
| 15363001001 | 14849201001 | 14033001001 | 01445604001 | 14359501001 |
| 15363002001 | 13776401001 | 12759301001 | 01445609001 | 15267901001 |
| 15616901001 | 14398601001 | 14148601001 | 01445605001 | |
| 00072601001 | 14398701001 | 14148501001 | 01445606001 | |
| 00072602001 | 15290001001 | 15603201001 | 01445607001 | |
| 00072603001 | 15868501001 | 13982501001 | 01445602001 | |
| 11725301001 | 13157101001 | 12734302001 | 01445603001 | |
| 11725302001 | 14404701001 | 12759102001 | 15960101001 | |
| 12881901001 | 14399701001 | 12689502001 | 12771001001 | |
| 14693401001 | 14399801001 | 13111502001 | 13947001001 | |
| 15440701001 | 15378701001 | 14040601001 | 07251001001 | |
| 15469801001 | 14847801001 | 12734301001 | 07339901001 | |
| 15470001001 | 12336401001 | 12759101001 | 09018701001 | |
| 15326101001 | 14848001001 | 14152701001 | 09018702001 | |
| 15892101001 | 14396301001 | 14165501001 | 14213701001 | |
| 15748501001 | 13826001001 | 14053001001 | 14031901001 | |
| 15892101001 | 14400001001 | 13109601001 | 13981601001 | |
| 15400501001 | 14400002001 | 12689501001 | 14165301001 | |
| 14269001001 | 13840901001 | 13111501001 | 14055901001 | |
| 00816701001 | 15900001001 | 14228101001 | 14055902001 | |
| 06821701001 | 13696801001 | 14151501001 | 15334201001 | |
| 12751901001 | 14982301001 | 14279401001 | 15583201001 | |
| 12751902001 | 15578501001 | 14182701001 | 08745601001 | |
| 13389401001 | 14400101001 | 14031501001 | 14741401001 | |
| 13485001001 | 14400102001 | 14048101001 | 15325601001 | |
| 13633501001 | 14955501001 | 13111401001 | 01555208001 | |
| 13709401001 | 14400201001 | 14279402001 | 08290701001 | |

| Prohibited PREF<br>Codes | Prohibited PREF<br>Codes | Prohibited PREF<br>Codes | Prohibited PREF<br>Codes | Prohibited PREF<br>Codes |
|---|---|---|---|---|
| 13769601001 | 14400202001 | 14216301001 | 14194301001 | |
| 13769901001 | 15502802001 | 13110601001 | 15269501001 | |
| 13770201001 | 15502801001 | 13111503001 | 14410101001 | |
| 13770901001 | 14400301001 | 13981901001 | 14183101001 | |
| 13771401001 | 14400302001 | 13982601001 | 14039401001 | |
| 13772801001 | 15868401001 | 13110701001 | 13980401001 | |
| 15464401001 | 01402505001 | 13110702001 | 01555209001 | |
| 01612901001 | 01612906001 | 14000501001 | 15500901001 | |
| 01612904001 | 01555204001 | 14030001001 | 15261201001 | |
| 01612903001 | 14193001001 | 14023901001 | 07872901001 | |
| 01612907001 | 14054001001 | 14034301001 | 15520801001 | |
| 01612911001 | 14054801001 | 15927901001 | 15539901001 | |
| 01612902001 | 14181501001 | 13980101001 | 15578201001 | |
| 01612909001 | 12759202001 | 14032301001 | 15628001001 | |
| 01612910001 | 14666301001 | 14032501001 | 15536601001 | |
| 01612905001 | 14000401001 | 15388901001 | 07252301001 | |
| 01612908001 | 12759201001 | 14407901001 | 01601501001 | |
| 14022001001 | 14032001001 | 14997401001 | 14972001001 | |
| 14156901001 | 14032401001 | 14151801001 | 13978201001 | |
| 14149701001 | 15632601001 | 13979301001 | 15586901001 | |

# 36) Hypersensitivity including Infusion-Related Reaction includes MedDRA Terms (MedDRA 25.0) listed in the following table:

| MedDRA Term Name | MedDRA Term Name | MedDRA Term Name | MedDRA Term Name |
|---|---|---|---|
| Acquired C1 inhibitor deficiency | Cross sensitivity reaction | Injection site urticaria | Skin necrosis |
| Acute generalised exanthematous pustulosis | Cutaneous vasculitis | Injection site vasculitis | Skin reaction |
| Administration related reaction | Dennie-Morgan fold | Instillation site hypersensitivity | Skin test positive |
| Administration site dermatitis | Dermal filler reaction | Instillation site rash | Solar urticaria |
| Administration site eczema | Dermatitis | Instillation site urticaria | Solvent sensitivity |

| MedDRA Term Name | MedDRA Term Name | MedDRA Term Name | MedDRA Term Name |
|---|---|---|---|
| Administration site hypersensitivity | Dermatitis acneiform | Interstitial granulomatous dermatitis | Stevens-Johnson syndrome |
| Administration site rash | Dermatitis allergic | Intestinal angioedema | Stoma site hypersensitivity |
| Administration site recall reaction | Dermatitis atopic | Iodine allergy | Stoma site rash |
| Administration site urticaria | Dermatitis bullous | Kounis syndrome | Stridor |
| Administration site vasculitis | Dermatitis contact | Laryngeal oedema | Swelling face |
| Allergic bronchitis | Dermatitis exfoliative | Laryngitis allergic | Swelling of eyelid |
| Allergic colitis | Dermatitis exfoliative generalised | Laryngospasm | Swollen tongue |
| Allergic cough | Dermatitis herpetiformis | Laryngotracheal oedema | Symmetrical drug-related intertriginous and flexural exanthema |
| Allergic cystitis | Dermatitis infected | Limbal swelling | Throat tightness |
| Allergic eosinophilia | Dermatitis psoriasiform | Lip oedema | Tongue oedema |
| Allergic gastroenteritis | Device allergy | Lip swelling | Toxic epidermal necrolysis |
| Allergic hepatitis | Dialysis membrane reaction | Mast cell activation syndrome | Toxic skin eruption |
| Allergic keratitis | Distributive shock | Mast cell degranulation present | Tracheal oedema |
| Allergic lymphangitis | Documented hypersensitivity to administered product | Medical device site dermatitis | Type I hypersensitivity |
| Allergic oedema | Drug eruption | Medical device site eczema | Type II hypersensitivity |
| Allergic otitis externa | Drug hypersensitivity | Medical device site hypersensitivity | Type III immune complex mediated reaction |
| Allergic otitis media | Drug provocation test | Medical device site rash | Type IV hypersensitivity reaction |
| Allergic pharyngitis | Drug reaction with eosinophilia and systemic symptoms | Medical device site recall reaction | Urticaria |
| Allergic reaction to excipient | Eczema | Medical device site urticaria | Urticaria cholinergic |
| Allergic respiratory disease | Eczema infantile | Mouth swelling | Urticaria chronic |

| MedDRA Term Name | MedDRA Term Name | MedDRA Term Name | MedDRA Term Name |
|---|---|---|---|
| Allergic respiratory symptom | Eczema nummular | Mucocutaneous rash | Urticaria contact |
| Allergic sinusitis | Eczema vaccinatum | Multiple allergies | Urticaria papular |
| Allergic stomatitis | Eczema vesicular | Nephritis allergic | Urticaria physical |
| Allergic transfusion reaction | Eczema weeping | Nikolsky's sign | Urticaria pigmentosa |
| Allergy alert test positive | Encephalitis allergic | Nodular rash | Urticaria vesiculosa |
| Allergy test positive | Encephalopathy allergic | Nutritional supplement allergy | Urticarial dermatitis |
| Allergy to immunoglobulin therapy | Eosinophilic<br>granulomatosis with<br>polyangiitis | Oculomucocutaneous syndrome | Urticarial vasculitis |
| Allergy to surgical sutures | Epidermal necrosis | Oculorespiratory syndrome | Vaccination site dermatitis |
| Allergy to vaccine | Epidermolysis | Oedema mouth | Vaccination site eczema |
| Anal eczema | Epidermolysis bullosa | Oral allergy syndrome | Vaccination site exfoliation |
| Anaphylactic reaction | Epiglottic oedema | Orbital swelling | Vaccination site hypersensitivity |
| Anaphylactic shock | Erythema multiforme | Oropharyngeal blistering | Vaccination site rash |
| Anaphylactic transfusion reaction | Erythema nodosum | Oropharyngeal oedema | Vaccination site recall reaction |
| Anaphylactoid reaction | Exfoliative rash | Oropharyngeal spasm | Vaccination site urticaria |
| Anaphylactoid shock | Eye allergy | Oropharyngeal swelling | Vaccination site vasculitis |
| Anaphylaxis treatment | Eye oedema | Palatal oedema | Vaccination site vesicles |
| Angioedema | Eye swelling | Palatal swelling | Vaginal ulceration |
| Anti-neutrophil cytoplasmic antibody positive vasculitis | Eyelid oedema | Palisaded neutrophilic granulomatous dermatitis | Vancomycin infusion reaction |
| Antiallergic therapy | Face oedema | Palpable purpura | Vascular access site dermatitis |
| Antiendomysial antibody positive | Fixed eruption | Pathergy reaction | Vascular access site eczema |
| Application site dermatitis | Flushing | Perioral dermatitis | Vasculitic rash |
| Application site eczema | Generalised bullous fixed drug eruption | Periorbital dermatitis | Vasodilatation |
| Application site hypersensitivity | Giant papillary conjunctivitis | Periorbital oedema | Vernal keratoconjunctivitis |
| Application site rash | Gingival oedema | Periorbital swelling | Vessel puncture site rash |

| MedDRA Term Name | MedDRA Term Name | MedDRA Term Name | MedDRA Term Name |
|---|---|---|---|
| Application site recall reaction | Gingival swelling | Pharyngeal oedema | Vessel puncture site vesicles |
| Application site urticaria | Gleich's syndrome | Pharyngeal swelling | Vulval eczema |
| Application site vasculitis | Haemorrhagic urticaria | Polymers allergy | Vulval ulceration |
| Arthritis allergic | Hand dermatitis | Post procedural fever | Vulvovaginal rash |
| Aspirin-exacerbated respiratory disease | Heart rate decreased | Procedural shock | Vulvovaginal ulceration |
| Atopic cough | Henoch-Schonlein purpura | Pruritus allergic | Vulvovaginitis allergic |
| Atopy | Henoch-Schonlein purpura nephritis | Pseudoallergic reaction | |
| Blepharitis allergic | Heparin-induced thrombocytopenia | Radioallergosorbent test positive | |
| Blood immunoglobulin E<br>abnormal | Hyperhidrosis | Rash | |
| Blood immunoglobulin E increased | Hypersensitivity | Rash erythematous | |
| Blood pressure decreased | Hypersensitivity myocarditis | Rash follicular | |
| Blood pressure diastolic decreased | Hypersensitivity pneumonitis | Rash macular | |
| Blood pressure diastolic increased | Hypersensitivity vasculitis | Rash maculo-papular | |
| Blood pressure increased | Hypertension | Rash maculovesicular | |
| Blood pressure systolic decreased | Hypotension | Rash morbilliform | |
| Blood pressure systolic increased | Idiopathic urticaria | Rash neonatal | |
| Bone cement allergy | Immediate post-injection reaction | Rash papulosquamous | |
| Bradyarrhythmia | Immune thrombocytopenia | Rash pruritic | |
| Bradycardia | Immune tolerance induction | Rash pustular | |
| Bromoderma | Implant site dermatitis | Rash rubelliform | |
| Bronchial obstruction | Implant site hypersensitivity | Rash scarlatiniform | |
| Bronchospasm | Implant site rash | Rash vesicular | |
| Bullous haemorrhagic dermatosis | Implant site urticaria | Reaction to azo-dyes | |

| MedDRA Term Name | MedDRA Term Name | MedDRA Term Name | MedDRA Term Name |
|---|---|---|---|
| Catheter site dermatitis | Incision site dermatitis | Reaction to colouring | |
| Catheter site eczema | Incision site rash | Reaction to excipient | |
| Catheter site hypersensitivity | Infusion related hypersensitivity reaction | Reaction to flavouring | |
| Catheter site rash | Infusion related reaction | Reaction to food additive | |
| Catheter site urticaria | Infusion site dermatitis | Reaction to preservatives | |
| Catheter site vasculitis | Infusion site eczema | Reaction to sweetener | |
| Chronic eosinophilic rhinosinusitis | Infusion site hypersensitivity | Rhinitis allergic | |
| Chronic hyperplastic eosinophilic sinusitis | Infusion site rash | Scleral oedema | |
| Circulatory collapse | Infusion site recall reaction | Scleritis allergic | |
| Circumoral oedema | Infusion site urticaria | Scrotal dermatitis | |
| Circumoral swelling | Infusion site vasculitis | Scrotal oedema | |
| Conjunctival oedema | Injection related reaction | Serum sickness | |
| Conjunctivitis allergic | Injection site dermatitis | Serum sickness-like reaction | |
| Contact stomatitis | Injection site eczema | Shock | |
| Contrast media allergy | Injection site hypersensitivity | Shock symptom | |
| Contrast media reaction | Injection site rash | Sinus bradycardia | |
| Corneal oedema | Injection site recall reaction | SJS-TEN overlap | |

# 37) COVID-19 vaccines include the following preferred term codes (WHODrug BMAR2022):

| <b>Prohibited PREF Codes</b> | <b>Prohibited PREF Codes</b> | Prohibited PREF Codes |
|---|---|---|
| 00002001001 | 15268629001 | 15268666001 |
| 06201402001 | 15268630001 | 15268667001 |
| 06439204001 | 15268631001 | 15268668001 |
| 06559301001 | 15268632001 | 15268669001 |
| 06559307001 | 15268633001 | 15268670001 |
| 13195801001 | 15268634001 | 15268671001 |
| 13949502001 | 15268635001 | 15268672001 |
| 13950013001 | 15268636001 | 15268673001 |

| <b>Prohibited PREF Codes</b> | Prohibited PREF Codes | Prohibited PREF Codes |
|------------------------------|-----------------------|-----------------------|
| 14953401001 | 15268637001 | 15268674001 |
| 14953501001 | 15268638001 | 15268675001 |
| 15092101001 | 15268639001 | 15268676001 |
| 15268601001 | 15268640001 | 15268677001 |
| 15268602001 | 15268641001 | 15268678001 |
| 15268603001 | 15268642001 | 15268679001 |
| 15268604001 | 15268643001 | 15268680001 |
| 15268605001 | 15268644001 | 15268681001 |
| 15268607001 | 15268645001 | 15268682001 |
| 15268609001 | 15268646001 | 15268683001 |
| 15268610001 | 15268647001 | 15268684001 |
| 15268611001 | 15268648001 | 15268685001 |
| 15268612001 | 15268649001 | 15268686001 |
| 15268613001 | 15268650001 | 15268687001 |
| 15268614001 | 15268651001 | 15268688001 |
| 15268615001 | 15268652001 | 15268689001 |
| 15268616001 | 15268653001 | 15268690001 |
| 15268617001 | 15268654001 | 15268691001 |
| 15268618001 | 15268655001 | 15268692001 |
| 15268619001 | 15268656001 | 15268693001 |
| 15268620001 | 15268657001 | 90031301001 |
| 15268621001 | 15268658001 | |
| 15268622001 | 15268659001 | |
| 15268623001 | 15268660001 | |
| 15268624001 | 15268661001 | |
| 15268625001 | 15268662001 | |
| 15268626001 | 15268663001 | |
| 15268627001 | 15268664001 | |
| 15268628001 | 15268665001 | |

# 38) Antithrombotic medications include the following drugs:

| Drug name |
|------------------------------------------------------|
| Direct factor Xa inhibitors |
| Direct thrombin inhibitors |
| Low molecular weight heparins (LMWH) and heparinoids |
| Other heparins |
| Other antithrombotic drugs |
| Platelet aggregation inhibitors, excluding heparin |
| Thrombolytic drugs |
| Vitamin K antagonists |
| Heparins |

# with preferred term codes (WHODrug BMAR2022):

| Prohibited<br>PREF Codes | Prohibited<br>PREF Codes | Prohibited<br>PREF Codes | Prohibited<br>PREF Codes | Prohibited<br>PREF Codes | Prohibited<br>PREF Codes | Prohibited<br>PREF Codes |
|---|---|---|---|---|---|---|
| 06259501001 | 13765501001 | 12384902001 | 12353501001 | 13595102001 | 11890502001 | 12800601001 |
| 06324201001 | 13765502001 | 13825101001 | 12353502001 | 11902101001 | 12829002001 | 11012901001 |
| 06324202001 | 13766301001 | 13825102001 | 12354601001 | 11902102001 | 12779502001 | 13576201001 |
| 06297801001 | 15159701001 | 13824801001 | 12354201001 | 12382602001 | 12779503001 | 11885501001 |
| 06297802001 | 15159702001 | 12385301001 | 12354202001 | 12382402001 | 12779602001 | 13576701001 |
| 06297803001 | 12430501001 | 12385501001 | 12353602001 | 12382601001 | 11485302001 | 90045701001 |
| 01551201001 | 12430502001 | 12384901001 | 12353601001 | 12382401001 | 11756602001 | 13185301001 |
| 01551202001 | 11096401001 | 13824501001 | 13623001001 | 12382403001 | 12150301001 | 12189002001 |
| 05705201001 | 11096402001 | 11549402001 | 12150502001 | 13749001001 | 11923801001 | 12189003001 |
| 01369401001 | 11902001001 | 11549401001 | 12150503001 | 13707401001 | 12151101001 | 12189001001 |
| 01369402001 | 11902002001 | 10534502001 | 12150501001 | 13707402001 | 11902401001 | 13599601001 |
| 01506801001 | 13600801001 | 10534501001 | 11610504001 | 11890503001 | 11641801001 | 13599602001 |
| 01506802001 | 12150602001 | 12268601001 | 11610502001 | 12406404001 | 13629501001 | 11442802001 |
| 01633201001 | 12150601001 | 12268602001 | 11610002001 | 12406403001 | 12150201001 | 11442801001 |
| 01633202001 | 01384201001 | 12269902001 | 11610203001 | 12382702001 | 11492701001 | 12180302001 |
| 01633203001 | 01384202001 | 12283302001 | 11610202001 | 11578403001 | 13313701001 | 12646902001 |
| 01288601001 | 11097102001 | 11177702001 | 14527702001 | 11578402001 | 12151401001 | 12646901001 |
| 01346001001 | 11678602001 | 12283301001 | 12406402001 | 11096101001 | 10907301001 | 00889601001 |
| 01384201001 | 11678601001 | 12269901001 | 12456903001 | 11096102001 | 11052701001 | 00889603001 |
| 01384202001 | 11097101001 | 11177701001 | 12456902001 | 12416702001 | 12286502001 | 00889602001 |
| 07368201001 | 13431901001 | 14427201001 | 12156601001 | 12416701001 | 12286501001 | 11866102001 |
| 07368202001 | 11623502001 | 14421501001 | 12156602001 | 00027701001 | 13572501001 | 11866101001 |
| 01708301001 | 11623501001 | 14488101001 | 11699802001 | 00027702001 | 12150701001 | 00723702001 |

| Prohibited | Prohibited | Prohibited | Prohibited | Prohibited | Prohibited | Prohibited |
|---|---|---|---|---|---|---|
| PREF Codes | PREF Codes | PREF Codes | PREF Codes | PREF Codes | PREF Codes | PREF Codes |
| 01708302001 | 13629801001 | 14488102001 | 11699803001 | 90006801001 | 12408701001 | 12344202001 |
| 01353901001 | 12181303001 | 01691801001 | 12186802001 | 00027705001 | 12406401001 | 11643102001 |
| 01353902001 | 12181302001 | 11699701001 | 11699602001 | 00027711001 | 12457201001 | 11012902001 |
| 06297801001 | 12181301001 | 11699702001 | 11699801001 | 00027710001 | 12456901001 | 13576202001 |
| 06297802001 | 07368201001 | 12475602001 | 12186801001 | 00027704001 | 12690401001 | 11885502001 |
| 06297803001 | 07368202001 | 12475601001 | 11699601001 | 00027708001 | 10999501001 | 01437701001 |
| 01707901001 | 12472001001 | 11375501001 | 14440702001 | 00027712001 | 12150901001 | 01437702001 |
| 01707902001 | 12472002001 | 11375502001 | 14440701001 | 00027707001 | 12382701001 | 07957701001 |
| 07957501001 | 11645802001 | 15876401001 | 01708201001 | 12150302001 | 12151201001 | 07957702001 |
| 07957502001 | 11645801001 | 15260602001 | 01708202001 | 11923802001 | 15778101001 | 00552101001 |
| 10679802001 | 10995602001 | 15260601001 | 12231802001 | 12151102001 | 12748001001 | 00552102001 |
| 13575901001 | 10995601001 | 12424001001 | 12231801001 | 11902402001 | 12517101001 | 11196102001 |
| 13575902001 | 12747502001 | 12424002001 | 11095802001 | 11641802001 | 11890501001 | 11657802001 |
| 10679801001 | 12747501001 | 10685602001 | 11095801001 | 13629502001 | 12829001001 | 11173402001 |
| 12601302001 | 12471001001 | 10685601001 | 11610503001 | 12150202001 | 14455101001 | 11196101001 |
| 12150802001 | 12471002001 | 01708301001 | 13472301001 | 11492702001 | 12779501001 | 11657801001 |
| 12150801001 | 11645702001 | 01708302001 | 13472302001 | 12151402001 | 12779601001 | 11173401001 |
| 12669701001 | 11645701001 | 01353901001 | 11718202001 | 10907302001 | 11485301001 | 13178201001 |
| 12669702001 | 11729402001 | 01353902001 | 11718201001 | 10907303001 | 15876301001 | 05509001001 |
| 11681801001 | 11729401001 | 07957801001 | 11610501001 | 11052702001 | 15878201001 | 05509002001 |
| 11681802001 | 12385504001 | 07957802001 | 11610001001 | 12150702001 | 11756601001 | 08069601001 |
| 12601301001 | 12385602001 | 07368001001 | 11610201001 | 12408702001 | 00723701001 | 08069602001 |
| 12430802001 | 12385601001 | 12190302001 | 14527701001 | 12457202001 | 13599501001 | 07579101001 |
| 13802202001 | 12385002001 | 12190301001 | 12382902001 | 12690402001 | 13720001001 | 07579102001 |
| 12431002001 | 12385001001 | 11514301001 | 12382302001 | 10999502001 | 13313601001 | 08336301001 |
| 12431001001 | 12479901001 | 11514302001 | 11885902001 | 12150902001 | 12180301001 | 01486301001 |
| 12430801001 | 12479902001 | 11732402001 | 12382301001 | 12151202001 | 12188202001 | 01063701001 |
| 13802201001 | 12385502001 | 11732301001 | 12382901001 | 12748002001 | 12188201001 | 00027709001 |
| 13802203001 | 12385503001 | 11732302001 | 11885901001 | 12748003001 | 12344201001 | 06563401001 |
| 15767701001 | 12385302001 | 11732401001 | 13595301001 | 12517103001 | 11643101001 | 06563402001 |
| 15767702001 | 12384903001 | 12354602001 | 13595101001 | 12517102001 | 11578401001 | |
| 01707901001 | 00075201001 | 00007401001 | 00014801001 | 00014803001 | 00014804001 | |
| 01707902001 | 00723901001 | 00062601001 | 00014805001 | 00014802001 | 00393001001 | |

# 39) Figures:

For figures, for a time point where n (sample size) is <= 5, data will not be displayed at that time point in the figure, but all data will be included in the corresponding table summary.

# GS-US-540-5912-SAP-Final Analysis ELECTRONIC SIGNATURES

| Signed by | Meaning of Signature | Server Date<br>(dd-MMM-<br>yyyy hh:mm:ss) |
|---|---|---|
| PPD | Biostatistics eSigned | 26-Jul-2022<br>17:28:10 |
| PPD | Clinical Research eSigned | 27-Jul-2022<br>14:25:46 |